CLINICAL TRIAL: NCT00567190
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Efficacy and Safety of Pertuzumab + Trastuzumab + Docetaxel vs. Placebo + Trastuzumab + Docetaxel in Previously Untreated HER2-Positive Metastatic Breast Cancer
Brief Title: A Study to Evaluate Pertuzumab + Trastuzumab + Docetaxel vs. Placebo + Trastuzumab + Docetaxel in Previously Untreated HER2-Positive Metastatic Breast Cancer
Acronym: CLEOPATRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TOC4129g; WO20698 (Other: Hoffmann-La Roche); 2007-002997-72 (EudraCT Number)
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Results first posted 2012-09-13 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Herceptin; Breast cancer; MBC; Taxotere; HER2; HER2 positive breast cancer; HER2 + breast cancer; HER2-positive; HER2-positive metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pertuzumab + Trastuzumab + Docetaxel (Experimental): Participants randomized to this arm received pertuzumab 420 milligrams (mg) intravenously (IV) once every 3 weeks (q3w) and trastuzumab 6 milligrams per kilogram (mg/kg) IV q3w, plus docetaxel 75 milligrams per square metre of body surface (mg/m^2) IV q3w (for at least 6 cycles; 1 cycle was 21 days). After Cycle 6, continuation of docetaxel treatment was at the discretion of the participant and treating physician. Participants remained in the treatment phase of the study until investigator-assessed radiographic or clinical evidence of disease progression, unmanageable toxicity, or study termination and were followed for survival until death, loss to follow-up, withdrawal of consent, or study termination.
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Docetaxel
- Placebo + Trastuzumab + Docetaxel (Placebo Comparator): Participants randomized to this arm received placebo IV q3w and trastuzumab 6 mg/kg IV q3w, plus docetaxel 75 mg/m^2 IV q3w (for at least 6 cycles; 1 cycle was 21 days). After Cycle 6, continuation of docetaxel treatment was at the discretion of the participant and treating physician. Participants remained in the treatment phase of the study until investigator-assessed radiographic or clinical evidence of disease progression, unmanageable toxicity, or study termination and were followed for survival until death, loss to follow-up, withdrawal of consent, or study termination.
  Interventions: Drug: Placebo; Drug: Trastuzumab; Drug: Docetaxel

INTERVENTIONS:
Drug: Pertuzumab — Pertuzumab was administered as an intravenous (IV) loading dose of 840 milligrams (mg) q3w on Day 1 of Cycle 1 (1 Cycle length = 21 days), and 420 mg q3w on Day 1 of subsequent cycles until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.
  Other Names: Perjeta; RO4368451; RG1273
  Arms: Pertuzumab + Trastuzumab + Docetaxel
Drug: Placebo — Placebo (matching pertuzumab) was administered intravenously.
  Arms: Placebo + Trastuzumab + Docetaxel
Drug: Trastuzumab — Trastuzumab was administered as an IV loading dose of 8 milligrams per kilogram (mg/kg) q3w on Day 2 of Cycle 1 (1 Cycle length = 21 days), and 6 mg/kg q3w on Day 1 of subsequent cycles until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.
  Other Names: Herceptin
Drug: Docetaxel — Docetaxel was administered as an IV dose of 75 milligrams per square meter of body surface area (mg/m^2) q3w on Day 2 of Cycle 1 (1 Cycle length = 21 days), and 75 mg/m^2 (up to 100 mg/m^2 as per treating physician discretion) q3w on Day 1 of subsequent cycles until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination. On or prior to Cycle 6, docetaxel was only to be discontinued for progressive disease or unmanageable toxicity. After Cycle 6, continuation of docetaxel treatment was at the discretion of the participant and treating physician.
  Other Names: Taxotere

SUMMARY:
This study was a Phase III, randomized, double-blind, placebo-controlled, multicenter international clinical trial conducted to investigate the use of pertuzumab in combination with trastuzumab and docetaxel as first-line treatment for participants with human epidermal growth factor receptor 2 (HER2)-positive metastatic breast cancer (MBC). Participants could have received one prior hormonal treatment for MBC. Participants may have received systemic breast cancer treatment in the neo-adjuvant or adjuvant setting, provided that the participant had experienced a disease-free interval (DFI) of greater than or equal to (≥)12 months from completion of adjuvant systemic treatment (excluding hormonal therapy) to metastatic diagnosis. Participants may have received trastuzumab and/or a taxane during the neo-adjuvant or adjuvant treatment.

Participants were randomized in 1:1 ratio to receive either pertuzumab or placebo, along with trastuzumab and docetaxel once every 3 weeks (q3w), during the treatment phase of the study until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination. Participants in the Placebo arm were not allowed to receive open-label pertuzumab after discontinuation from study treatment. However, if any analysis of overall survival had met the predefined criteria for statistical significance, participants in the Placebo arm still on treatment were offered the option to receive open-label pertuzumab in addition to other study medications.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast with locally recurrent or metastatic disease, and candidate for chemotherapy. Participants with measurable and non-measurable disease are eligible (locally recurrent disease must not be amenable to resection with curative intent; participants with de novo Stage IV disease are eligible)
* Human epidermal growth factor receptor 2 (HER2)-positive metastatic breast cancer (MBC)
* Left ventricular ejection fraction (LVEF) ≥50 percent (%) at baseline (within 42 days of randomization)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* For women of childbearing potential and men with partners of childbearing potential, agreement to use a highly effective form of contraception and to continue its use for the duration of study treatment and for at least 7 months after the last dose of study treatment

Exclusion Criteria:

* History of anti-cancer therapy for MBC (with the exception of one prior hormonal regimen for MBC, which must be stopped prior to randomization)
* History of approved or investigative tyrosine kinase/HER inhibitors for breast cancer in any treatment setting, except trastuzumab used in the neoadjuvant or adjuvant setting
* History of systemic breast cancer treatment in the neo-adjuvant or adjuvant setting with a disease-free interval from completion of the systemic treatment (excluding hormonal therapy) to metastatic diagnosis of less than (<)12 months
* History of persistent Grade ≥2 hematologic toxicity resulting from previous adjuvant therapy
* Current peripheral neuropathy of National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 3.0, Grade ≥3 at randomization
* History of other malignancy within the last 5 years, except for carcinoma in situ of the cervix, basal cell carcinoma or squamous cell carcinoma of the skin that has been previously treated with curative intent
* Current clinical or radiographic evidence of central nervous system (CNS) metastases
* Computed tomography (CT) or magnetic resonance imaging (MRI) scan of the brain is mandatory in cases of clinical suspicion of brain metastases
* History of exposure to cumulative doses of anthracyclines
* Current uncontrolled hypertension or unstable angina
* History of congestive heart failure (CHF) of any New York Heart Association (NYHA) criteria, or serious cardiac arrhythmia requiring treatment (exception: atrial fibrillation or paroxysmal supraventricular tachycardia)
* History of myocardial infarction within 6 months of randomization
* History of LVEF decline to below 50% during or after prior trastuzumab neo-adjuvant or adjuvant therapy
* Current dyspnea at rest due to complications of advanced malignancy, or other diseases that require continuous oxygen therapy
* Inadequate organ function, as defined in the protocol, within 28 days prior to randomization
* Current severe, uncontrolled systemic disease
* Major surgical procedure or significant traumatic injury within 28 days prior to study treatment start or anticipation of the need for major surgery during the course of study treatment
* Pregnant or lactating women
* History of receiving any investigational treatment within 28 days of randomization
* Current known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)
* Receipt of IV antibiotics for infection within 14 days of randomization
* Current chronic daily treatment with corticosteroids (excluding inhaled steroids)
* Known hypersensitivity to any of the study drugs
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 2008-02-12 (Actual); Primary Completion 2011-05-13 (Actual); Study Completion 2018-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc./Hoffmann-La Roche
Locations (322):
- United States (159):
  - HonorHealth Research Institute - Bisgrove, Scottsdale, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Central Hematology Oncology Medical Group Inc., Alhambra, California
  - Pacific Cancer Medical Center, Anaheim, California
  - Comprehensive Blood/Cancer Ctr, Bakersfield, California
  - Kaiser Permanente - Baldwin Park, Baldwin Park, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - South Bay Oncology Hematology Partners, Campbell, California
  - Wilshire Oncology Medical Group, Corona, California
  - Compassionate Cancer Care, Fountain Valley, California
  - Pacific Coast Hematology/Oncology Medical Group, Fountain Valley, California
  - St. Jude Heritage Healthcare; Virgiia K.Crosson Can Ctr, Fullerton, California
  - Wilshire Onc Med Grp., Inc, Glendora, California
  - Wilshire Oncology Medical Group, La Verne, California
  - UCLA, Los Angeles, California
  - LAC USC Medical Center, Los Angeles, California
  - Cedars- Sinai Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center Clin Lab, Los Angeles, California
  - TORI Central Administration, Los Angeles, California
  - UCLA Hematology / Oncology Clinic, Los Angeles, California
  - UCLA Med Ctr; Pharma Svcs, Los Angeles, California
  - Sutter Gould Medical Foundation; Clinical Research, Modesto, California
  - Kaiser Permanente - Oakland, Oakland, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - UCLA Healthcare/Pasadena Oncology, Pasadena, California
  - Wilshire Oncology Medical Group, Pasadena, California
  - Bay Area Cancer Research Group, LLC, Pleasant Hill, California
  - Wilshire Oncology Medical Group, Pomona, California
  - Wilshire Oncology Medical Group, Rancho Cucamonga, California
  - UC Davis Cancer Center; Oncology, Sacramento, California
  - Kaiser Permanente San Diego; Hepatology Research, San Diego, California
  - K. Permanente - San Fransisco, San Francisco, California
  - K. Permanente - San Jose, San Jose, California
  - Sansum Santa Barbara Medical Foundation Clinic, Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - UCLA Hematology/Oncology, Santa Monica, California
  - UCLA / Santa Clarita Valley Cancer Center, Valencia, California
  - Kaiser Permanente - Vallejo, Vallejo, California
  - K. Permanente - Walnut Creek, Walnut Creek, California
  - Wilshire Oncology Medical Group, West Covina, California
  - Innovative clinical research institute/American institute of research, Whittier, California
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - MedStar Washington Hosp Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Boca Raton Comprehensive Cancer Center, Boca Raton, Florida
  - Florida Cancer Specialists -Cape Coral (Cape Coral Pkwy), Cape Coral, Florida
  - Florida Cancer Specialists - Cape Coral (Del Prado Blvd), Cape Coral, Florida
  - Northwest Oncology/ Hematology Assoc., Coral Springs, Florida
  - UM Sylvester Deerfield Beach; Sylvester Cancer Ctr, Deerfield Beach, Florida
  - Florida Cancer Specialists - Englewood, Englewood, Florida
  - Florida Cancer Specialists - Fort Myers (New Hampshire Ct), Fort Myers, Florida
  - Florida Cancer Specialists - Broadway, Fort Myers, Florida
  - Florida Cancer Specialists; SCRI, Fort Myers, Florida
  - Florida Cancer Specialists-Broadway, Fort Myers, Fort Myers, Florida
  - Private Practice Robert R. Carroll, Md, Pa, Gainesville, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Florida Cancer Specialists - Goodlette, Naples, Naples, Florida
  - Florida Cancer Specialists - Pine Ridge, Naples, Naples, Florida
  - Private Practice, Orlando, Florida
  - Breast Cancer Centre at Memorial Hospital West, Pembroke Pines, Florida
  - Florida Cancer Specialists - Port Charlotte, Port Charlotte, Florida
  - Florida Cancer Specialists; Sarasota, Sarasota, Florida
  - Bay Area Oncology, Tampa, Florida
  - Florida Cancer Specialists - Venice (S. Tamiami Tr), Venice, Florida
  - Florida Cancer Specialists - Sunset Lake, Venice, Venice, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Northeast Georgia Medical Center; Oncology Research Dept-5C, Gainesville, Georgia
  - Central Georgia Hematology Oncology Associates, Macon, Georgia
  - Northwest Georgia Oncology Centers, a Service of WellStar Cobb Hospital, Marietta, Georgia
  - Central GA Cancer Care, Warner Robins, Georgia
  - Elmhurst Hospital, Elmhurst, Illinois
  - Hematology Oncology Consultants Ltd, Naperville, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Midwestern Regional Medical Center; Office of Research, Zion, Illinois
  - Monroe Medical Associates - Hobart, Hobart, Indiana
  - St. Mary Medical Center, Hobart, Indiana
  - Hematology-Oncology of Indiana, Pc, Indianapolis, Indiana
  - Community Hospital; Pharmacy, Munster, Indiana
  - Northwest Oncology, Munster, Indiana
  - Monroe Medical Associates, Munster, Indiana
  - Family Medicine Vincennes, Vincennes, Indiana
  - Uni of Iowa Hospital&Clinic; Holden Comprehens. Cancer Ctr, Iowa City, Iowa
  - University of Kansas; Medical Center & Medical pavilion, Westwood, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Jewish Cancer Care, Louisville, Kentucky
  - Cancer Center of Acadiana at Lafayette General, Lafayette, Louisiana
  - Christus Schumpert Health System, Shreveport, Louisiana
  - Private Practice- Carolyn Hendricks, MD, Bethesda, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Berkshire Hematology, Oncology Pc, Pittsfield, Massachusetts
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Cancer & Hematology Center of West Michigan, Grand Rapids, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Southdale Cancer Clinic U of M Medical Center, Fairview- Edina, Edina, Minnesota
  - US Oncology Research at Minnesota Oncology, Minneapolis, Minnesota
  - Minneapolis Oncology Hamatology PA, Minneapolis, Minnesota
  - The Jones Clinic, PC, New Albany, Mississippi
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Southeast Nebraska Cancer Center;; Southeast Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Norfolk Oncology Consultants, Norfolk, Nebraska
  - Hematology-Oncology Consultants, Pc, Omaha, Nebraska
  - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - St. Barnabas Cancer Center, Livingston, New Jersey
  - Oncology and Hematology Specialists, Mountain Lakes, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Brockport-Interlakes Foundation, Brockport, New York
  - Canandaigua-Interlakes Found, Canandaigua, New York
  - Geneva-Interlakes Foundation, Geneva, New York
  - ProHEALTH Care Associates LLP, Lake Success, New York
  - Beth Israel Comprehensive Cancer Center Pharmacy, New York, New York
  - The Women'sOncology & Wellness Practice, New York, New York
  - Upstate Ny Cancer Research & Education Foundation, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Carolina Oncology Specialists, PA - Hickory, Hickory, North Carolina
  - Carolina BioOncology Institute, PLCC, Huntersville, North Carolina
  - NW Carolina Onc & Hem, Lenoir, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Hema Onc Conslts-Grant Ave, Columbus, Ohio
  - The Mark H. Zangmeister Ctr; Mid Ohio Onc/Hem Inc., Columbus, Ohio
  - Hematology Onc Consultants, Columbus, Ohio
  - Gabrail Cancer Center, Dover, Ohio
  - Hematology Oncology Consultants (NWK), Granville, Ohio
  - Medical College of Ohio; Cancer Institute, Toledo, Ohio
  - Mercy Physicians of Oklahoma, Oklahoma City, Oklahoma
  - CA Care Associates-OK Oncology and Hematology, Tulsa, Oklahoma
  - Cancer Care Assoc-S. Ingo, Tulsa, Oklahoma
  - OK Oncology & Hematology PC, Tulsa, Oklahoma
  - Cons in Med Onc and Hem, Darby, Pennsylvania
  - Consultants in Medical Oncology/Hematology, Drexel Hill, Pennsylvania
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania
  - Conslts in Med Onc (Newtown); Bryn Mawr Health Canc Ctr, Newtown Square, Pennsylvania
  - Uni of Pittsburgh; Magee-Women'S Hospital, Pittsburgh, Pennsylvania
  - Consultants Med Onc & Hem, Ridley Park, Pennsylvania
  - Erlanger Health System; Oncology Research, Chattanooga, Tennessee
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - McLeod Cancer and Blood Center, Johnson City, Tennessee
  - University of Tennessee Cancer Institute;Hem-Onc Consultants, Knoxville, Tennessee
  - Sarah Cannon Cancer Center - Tennessee Oncology, Pllc, Nashville, Tennessee
  - Park Plaza, Houston, Texas
  - Southwest, Houston, Texas
  - St. Joseph's, Houston, Texas
  - Memorial City-Main Office, Houston, Texas
  - Oncology Consultants, Houston, Texas
  - St. Luke's, Houston, Texas
  - Willowbrook, Houston, Texas
  - Katy-Christus St. Catherine, Katy, Texas
  - South Texas Oncology Hematology, San Antonio, Texas
  - Oncology Consultants - Sugar Land, Sugar Land, Texas
  - Northern Utah Associates, Ogden, Utah
  - Community Cancer Center Rutland Regional Medical Center, Rutland, Vermont
  - Wellmonth Physician Services, Bristol, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
  - St. Mary Medical Center, Walla Walla, Washington
- Argentina (7):
  - Sanatorio Güemes; Oncología, Buenos Aires
  - Centro de Oncologia e Investigacion Buenos Aires (COIBA), Buenos Aires
  - Instituto Medico Especializado (IME); Oncologia, Caba
  - Center Instituto Médico Privado I.M.P.; Oncology, Chaco-resistencia
  - Policlinica Privada Site la Plata SA; Oncology, La Plata
  - Unidad Oncológica De Neuquén, Neuquén
  - Hosp Provincial D. Centenarios; Oncology Dept, Rosario
- Brazil (19):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Clinica Amo - Assistencia Medica Em Oncologia, Salvador, Estado de Bahia
  - Centro Goiano de Oncologia - CGO, Goiânia, Goiás
  - Instituto Nacional de Cancer - INCa; Oncologia, Rio de Janeiro, Rio de Janeiro
  - Hospital Universitario Clementino Fraga Filho - UFRJ; Oncologia, Rio de Janeiro, Rio de Janeiro
  - Hospital de Caridade de Ijui; Oncologia, Ijuí, Rio Grande do Sul
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Hospital das Clinicas - FMUSP Ribeirao Preto, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC - FMABC; Oncologia e Hematologia, Santo André, São Paulo
  - Iso - Inst. Santista de Oncologia, Santos, São Paulo
  - Instituto do Cancer Arnaldo Vieira de Carvalho - ICAVC; Pesquisa Clinica, São Paulo, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Perola Byington, São Paulo, São Paulo
  - Inst. Brasileiro de Controle Ao Cancer; Oncologia Clinica / Quimioterapia, São Paulo, São Paulo
  - Hospital Estadual do Servidor Publico, São Paulo, São Paulo
  - Instituto de Oncologia de Sorocaba - CEPOS, Sorocaba, São Paulo
- St. Michael'S Hospital, Toronto, Ontario, Canada
- China (5):
  - Jilin Cancer Hospital, Changchun
  - Fuzhou General Hospital, PLA Nanjing Military Area Command, Fuzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Shanghai First People's Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
- Hospital Cima San Jose; Oncology, San José, Costa Rica
- Croatia (2):
  - Clinical Hospital Sisters of Mercy, Zagreb
  - University Hospital Centre Zagreb; Clinic For Oncology, Zagreb
- Ecuador (4):
  - Solca Guayaquil- Sociedad de Lucha Contra El Cáncer; Oncology, Guayaquil
  - Teodoro Maldonado Carbo Hospital; Oncology Service, Guayaquil
  - Hospital Carlos Andrade Marin; Servicio de Oncología, Quito
  - Hospital Solca Quito; Oncologia, Quito
- Finland (2):
  - Tampere University Hospital; Dept of Oncology, Tampere
  - Turku Uni Central Hospital; Oncology Clinics, Turku
- France (8):
  - Centre Oncologie Du Pays Basque, Bayonne
  - Clinique Tivoli; Sce Radiotherapie, Bordeaux
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - Centre Hospitalier Departemental Les Oudairies, La Roche-sur-Yon
  - Centre Jean Bernard, Le Mans
  - Centre Antoine Lacassagne; Hopital De Jour A2, Nice
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
  - Groupe Hospitalier Sud; Oncologie Radiotherapie, Salouël
- Germany (13):
  - Onkologischer Schwerpunkt am Oskar-Helene-Heim; Dres. Herrenberger, Keitel-Wittig u. Kirsch, Berlin
  - Onkologische Schwerpunktpraxis Bielefeld; Haemotologie & Internistische onkologie, Bielefeld
  - St. Elisabeth Krankenhaus Köln GmbH; Gynäkologie und Geburtshilfe, Cologne
  - Universitätsklinikum Essen; Zentrum Für Frauenheilkunde, Essen
  - Universitätsklinikum Halle (Saale); Universitätsklinik Und Poliklinik Für Gynäkologie, Halle
  - Universitätsklinikum Hamburg-Eppendorf; Frauenklinik, Hamburg
  - Nationales Centrum für Tumorerkrankungen (NCT) ; Gyn. Onk. Frauenklinik; Uniklinikum Heidelberg, Heidelberg
  - Universitätsmedizin Mainz; Klinik u. Poliklinik f. Geburtshilfe u. Frauenheilkunde, Mainz
  - Krankenhaus Rheinfelden; Frauenklinik, Rheinfelden
  - Robert-Bosch-Krankenhaus; Hämatologie, Onkologie und Palliativmedizin, Stuttgart
  - Klinikum Mutterhaus der Borromaeerinnen gGmbH; Haematologie/Onkologie, Trier
  - Universitätsklinik Tübingen; Frauenklinik, Tübingen
  - Haematologisch-Onkologische Praxis; Dr. med. Christoph Maintz und Matthias Groschek, Würselen
- Guatemala (3):
  - Centro Oncologico S.A., Guatemala City
  - Grupo Angeles, Guatemala City
  - Therapeutic Research Inst. & Lab S.A. (Trial), Guatemala City
- Hong Kong (2):
  - Pamela Youde Nethersole Eastern Hospital; Clinical Oncology, Hong Kong
  - Prince of Wales Hosp; Dept. Of Clinical Onc, Shatin
- Italy (10):
  - Policlinico Ospedaliero Ss Annunziata; U.O. Di Clinica Oncologica, Chieti, Abruzzo
  - Ospedale Antonio Perrino; Oncologia Medica, Brindisi, Apulia
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Ospedale Provinciale Santa Maria delle Croci, Ravenna, Emilia-Romagna
  - Ausl Frosinone - Ospedale Umberto I; Divisione Di Oncologia, Frosinone, Lazio
  - Az. Osp. Spedali Civili; Divisione Di Oncologia - Iii Medicina, Brescia, Lombardy
  - Fondazione Del Piemonte Per L'oncologia IRCC Di Candiolo, Candiolo, Piedmont
  - Ospedale Di Macerata; Oncologia, Macerata, The Marches
  - Azienda Sanitaria S. Maria Annunziata; S. C. Oncologia Medica, Antella (FI), Tuscany
  - Ospedale Misericordia E Dolce; Oncologia Medica, Prato, Tuscany
- Japan (28):
  - Aichi Cancer Center Hospital, Breast Oncology, Aichi
  - Chiba Cancer Center; Breast Surgical Oncology, Chiba
  - National Cancer Center Hospital East; Breast and Medical Oncology, Chiba
  - Natl Hosp Org Shikoku; Cancer Ctr, Surgery, Ehime
  - Kitakyushu Municipal Medical Center, Surgery, Fukuoka
  - National Hospital Organization Kyushu Cancer Center;Breast Oncology, Fukuoka
  - Gunma University Hospital; Department of Thoracic and Visceral Organ Surgery, Gunma
  - Sagara Hospital; Breast Surgery, Kagoshima
  - St. Marianna University School of Medicine Hospital, Breast and Endocrine Surgery, Kanagawa
  - Tokai University Hospital, Breast and Endocrine Surgery, Kanagawa
  - Kumamoto City Hospital, Breast and Endocrine Surgery, Kumamoto
  - Kumamoto Shinto General Hospital; Breast Cancer Center, Kumamoto
  - Kyoto University Hospital; Breast Surgery, Kyoto
  - Niigata Cancer Ctr Hospital; Breast Surgery, Niigata
  - Iwate Med Univ School of Med; Surgery, Numakunai
  - OSAKA CITY GENERAL HOSPITAL;Medical Oncology, Osaka
  - National Hospital Organization Osaka National Hospital; Breast Surgery, Osaka
  - Osaka University Hospital; Breast and Endocrine Surgery, Osaka
  - Saitama Medical University International Medical Center; Medical Oncology, Saitama
  - Saitama Cancer Center, Breast Oncology, Saitama
  - Shizuoka Cancer Center; Female Internal Medicine, Shizuoka
  - Shizuoka General Hospital; Breast Surgery, Shizuoka
  - Jichi Medical University; Dept of Clinical Oncology, Tochigi
  - National Cancer Center Hospital; Breast and Medical Oncology, Tokyo
  - St. Luke's Internat. Hospital, Breast Surgical Oncology, Tokyo
  - Tokyo Metropolitan; Komagome Hospital, Surgery, Tokyo
  - The Cancer Inst. Hosp. of JFCR; Breast Oncology Center, Tokyo
  - Tokyo Medical Uni. Hospital; Breast Oncology, Tokyo
- Latvia (3):
  - Daugavpils Regional Hospital, Daugavpils
  - Rigas Austrumu Kliniska Universitates slimnica, Latvijas Onkologijas centrs, Riga
  - P.Stradins Clinical University Hospital, Oncology Centre, Riga
- Mexico (2):
  - Hospital Angeles Metropolitano; Room 220, Mexico City, Mexico CITY (federal District)
  - Centro Oncologico Estatal ISSEMYM, Toluca
- North Macedonia (3):
  - Clinical Hospital; Oncology Department, Bitola
  - Institute of Radiotherapy Oncology, Skopje
  - Private Health Organization Acibadem Sistina Hospital, Skopje
- Philippines (3):
  - Cebu Cancer Institute; Perpetual Succour Hospital, Cebu City
  - Veterans Memorial Medical Center; Oncology, Quezon City
  - St Luke'S Medical Centre; Oncology, Quezon City
- Poland (5):
  - Samodzielny Publiczny Kliniczny Nr 1 W Lublinie; Klinika Chirurgii Onkologicznej, Lublin
  - COZL Oddzial Onkologii Klinicznej z pododdzialem Chemioterapii Dziennej, Lublin
  - Oddzial Chemioterapii Szpitala Klinicznego Nr 1 w Poznaniu, Poznan
  - Zachodniopomorskie Centrum Onkologii, Osrodek Innowacyjnosci, Rozwoju i Badan Klinicznych, Szczecin
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej-Curie Klinika Nowotworów Piersi i Chirurgii, Warsaw
- Russia (9):
  - FSBI"National Medical Research Center of Oncology named after N.N.Petrov" MHRF, Saint Petersburg, Sankt-Peterburg
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Regional Oncology Hospital Of Kursk; Chemotherapy, Kislino, Kursk Region
  - Blokhin Cancer Research Center; Combined Treatment, Moscow
  - Russian Oncology Research Center n.a. N.N. Blokhin Dpt of Clinical Pharmacology and Chemotherapy, Moscow
  - Omsk Region Clinical Oncology Dispensary; 1St Sergical Department, Omsk
  - State Inst. Of Healthcare Orenburg Regional Clinical Oncology Dis, Orenburg
  - SBI of Healthcare Leningrad Regional Oncology Dispensary, Saint Petersburg
  - SBI of Healthcare Samara Regional Clinical Oncology Dispensary, Samara
- Singapore (2):
  - National University Hospital; National University Cancer Institute, Singapore (NCIS), Singapore
  - National Cancer Centre; Medical Oncology, Singapore
- South Korea (5):
  - National Cancer Center; Medical Oncology, Gyeonggi-do
  - Seoul National Uni Hospital; Dept. of Internal Medicine/Hematology/Oncology, Seoul
  - Yonsei Uni College of Medicine, Severance Hospital; Internal Medicine Dept., Seoul
  - Samsung Medical Centre; Division of Hematology/Oncology, Seoul
  - Asan Medical Center, Uni Ulsan Collegemedicine; Dept.Internal Medicine / Divisionhematology/Oncology, Seoul
- Spain (9):
  - Hospital Universitario de Canarias;servicio de Oncologia, San Cristóbal de La Laguna, Tenerife
  - Complejo Hospitalario Universitario A Coruña (CHUAC, Materno Infantil), Oncología, A Coruña
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Duran i Reynals; Oncologia, Barcelona
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Hospital Universitari Arnau de Vilanova de Lleida; Servicio de Oncologia, Lleida
  - Centro Oncologico MD Anderson Internacional; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
- Thailand (6):
  - Chulalongkorn Hospital; Medical Oncology, Bangkok
  - National Cancer Inst., Bangkok
  - Rajavithi Hospital; Division of Medical Oncology, Bangkok
  - Ramathibodi Hospital; Dept of Med.-Div. of Med. Onc, Bangkok
  - Faculty of Med. Siriraj Hosp.; Med.-Div. of Med. Oncology, Bangkok
  - Songklanagarind Hospital; Department of Oncology, Songkhla
- United Kingdom (11):
  - Broomfield Hospital; Oncology, Chelmsford
  - St James Uni Hospital; Icrf Cancer Medicine Research Unit, Leeds
  - Leicester Royal Infirmary; Dept. of Medical Oncology, Leicester
  - St. Bartholomew'S Hospital; Dept of Medical Oncology, London
  - Royal Free Hospital; Dept of Oncology, London
  - St George'S Hospital; Oncology Research Office /Oncology Opd, London
  - Charing Cross Hospital; Medical Oncology., London
  - The Clatterbridge Cancer Ctr For Oncolgy, Metropolitan Borough of Wirral
  - Mount Vernon Hospital; Centre For Cancer Treatment, Northwood
  - Royal Cornwall Hospital; Dept of Clinical Oncology, Truro
  - Southend Hospital; Oncology Dept, Westcliffe-on-sea

REFERENCES:
- [Result] Baselga J, Cortes J, Kim SB, Im SA, Hegg R, Im YH, Roman L, Pedrini JL, Pienkowski T, Knott A, Clark E, Benyunes MC, Ross G, Swain SM; CLEOPATRA Study Group. Pertuzumab plus trastuzumab plus docetaxel for metastatic breast cancer. N Engl J Med. 2012 Jan 12;366(2):109-19. doi: 10.1056/NEJMoa1113216. Epub 2011 Dec 7. PMID 22149875
- [Derived] Swain SM, Miles D, Kim SB, Im YH, Im SA, Semiglazov V, Ciruelos E, Schneeweiss A, Loi S, Monturus E, Clark E, Knott A, Restuccia E, Benyunes MC, Cortes J; CLEOPATRA study group. Pertuzumab, trastuzumab, and docetaxel for HER2-positive metastatic breast cancer (CLEOPATRA): end-of-study results from a double-blind, randomised, placebo-controlled, phase 3 study. Lancet Oncol. 2020 Apr;21(4):519-530. doi: 10.1016/S1470-2045(19)30863-0. Epub 2020 Mar 12. PMID 32171426
- [Derived] Miles D, Im YH, Fung A, Yoo B, Knott A, Heeson S, Beattie MS, Swain SM. Effect of docetaxel duration on clinical outcomes: exploratory analysis of CLEOPATRA, a phase III randomized controlled trial. Ann Oncol. 2017 Nov 1;28(11):2761-2767. doi: 10.1093/annonc/mdx406. PMID 29112701
- [Derived] Swain SM, Schneeweiss A, Gianni L, Gao JJ, Stein A, Waldron-Lynch M, Heeson S, Beattie MS, Yoo B, Cortes J, Baselga J. Incidence and management of diarrhea in patients with HER2-positive breast cancer treated with pertuzumab. Ann Oncol. 2017 Apr 1;28(4):761-768. doi: 10.1093/annonc/mdw695. PMID 28057664
- [Derived] Luen SJ, Salgado R, Fox S, Savas P, Eng-Wong J, Clark E, Kiermaier A, Swain SM, Baselga J, Michiels S, Loi S. Tumour-infiltrating lymphocytes in advanced HER2-positive breast cancer treated with pertuzumab or placebo in addition to trastuzumab and docetaxel: a retrospective analysis of the CLEOPATRA study. Lancet Oncol. 2017 Jan;18(1):52-62. doi: 10.1016/S1470-2045(16)30631-3. Epub 2016 Dec 7. PMID 27964843
- [Derived] Swain SM, Baselga J, Kim SB, Ro J, Semiglazov V, Campone M, Ciruelos E, Ferrero JM, Schneeweiss A, Heeson S, Clark E, Ross G, Benyunes MC, Cortes J; CLEOPATRA Study Group. Pertuzumab, trastuzumab, and docetaxel in HER2-positive metastatic breast cancer. N Engl J Med. 2015 Feb 19;372(8):724-34. doi: 10.1056/NEJMoa1413513. PMID 25693012
- [Derived] Baselga J, Cortes J, Im SA, Clark E, Ross G, Kiermaier A, Swain SM. Biomarker analyses in CLEOPATRA: a phase III, placebo-controlled study of pertuzumab in human epidermal growth factor receptor 2-positive, first-line metastatic breast cancer. J Clin Oncol. 2014 Nov 20;32(33):3753-61. doi: 10.1200/JCO.2013.54.5384. Epub 2014 Oct 20. PMID 25332247
- [Derived] Swain SM, Baselga J, Miles D, Im YH, Quah C, Lee LF, Cortes J. Incidence of central nervous system metastases in patients with HER2-positive metastatic breast cancer treated with pertuzumab, trastuzumab, and docetaxel: results from the randomized phase III study CLEOPATRA. Ann Oncol. 2014 Jun;25(6):1116-21. doi: 10.1093/annonc/mdu133. Epub 2014 Mar 31. PMID 24685829
- [Derived] Miles D, Baselga J, Amadori D, Sunpaweravong P, Semiglazov V, Knott A, Clark E, Ross G, Swain SM. Treatment of older patients with HER2-positive metastatic breast cancer with pertuzumab, trastuzumab, and docetaxel: subgroup analyses from a randomized, double-blind, placebo-controlled phase III trial (CLEOPATRA). Breast Cancer Res Treat. 2013 Nov;142(1):89-99. doi: 10.1007/s10549-013-2710-z. Epub 2013 Oct 16. PMID 24129974
- [Derived] Cortes J, Baselga J, Im YH, Im SA, Pivot X, Ross G, Clark E, Knott A, Swain SM. Health-related quality-of-life assessment in CLEOPATRA, a phase III study combining pertuzumab with trastuzumab and docetaxel in metastatic breast cancer. Ann Oncol. 2013 Oct;24(10):2630-2635. doi: 10.1093/annonc/mdt274. Epub 2013 Jul 17. PMID 23868905
- [Derived] Swain SM, Kim SB, Cortes J, Ro J, Semiglazov V, Campone M, Ciruelos E, Ferrero JM, Schneeweiss A, Knott A, Clark E, Ross G, Benyunes MC, Baselga J. Pertuzumab, trastuzumab, and docetaxel for HER2-positive metastatic breast cancer (CLEOPATRA study): overall survival results from a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Oncol. 2013 May;14(6):461-71. doi: 10.1016/S1470-2045(13)70130-X. Epub 2013 Apr 18. PMID 23602601
- [Derived] Baselga J, Swain SM. CLEOPATRA: a phase III evaluation of pertuzumab and trastuzumab for HER2-positive metastatic breast cancer. Clin Breast Cancer. 2010 Dec 1;10(6):489-91. doi: 10.3816/CBC.2010.n.065. PMID 21147694

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1196 patients were screened for the study, of whom a total of 808 participants were randomized to one of the two treatment arms.
Period: Overall Study
Arm/Group | Pertuzumab + Trastuzumab + Docetaxel | Placebo + Trastuzumab + Docetaxel
Started (Intent-to-Treat (ITT) Population) | 402 | 406
Did Not Receive Any Study Treatment | 2 | 2
Received at Least One Dose of Pertuzumab (Safety Population (Pertuzumab)) | 399 | 9 (9 participants randomized to the Placebo arm actually received at least one dose of pertuzumab.)
Received at Least One Dose of Placebo (Safety Population (Placebo)) | 1 (1 participant randomized to the Pertuzumab arm actually received placebo at every treatment cycle.) | 395
Crossover From Placebo to Pertuzumab | 0 | 50 (From July 2012, 50 participants randomized to Placebo arm crossed over to open-label pertuzumab.)
Completed (Alive and in Survival Follow-up at End of Study) | 119 | 73
Not Completed | 283 | 333
Not completed — Death | 235 | 280
Not completed — Withdrew Consent or Lost to Follow-up | 48 | 53

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Pertuzumab + Trastuzumab + Docetaxel | Placebo + Trastuzumab + Docetaxel | Total
Number analyzed (Participants) | 402 | 406 | 808
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (10.94) | 53.5 (11.35) | 53.5 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 402 | 404 | 806
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 44 | 83
  Not Hispanic or Latino | 362 | 362 | 724
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 128 | 133 | 261
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 20 | 30
  White | 245 | 235 | 480
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 14 | 30
Region [Count of Participants; unit: Participants]
  Asia | 125 | 128 | 253
  Europe | 154 | 152 | 306
  North America | 67 | 68 | 135
  South America | 56 | 58 | 114
Prior Treatment Status [Count of Participants; unit: Participants]
  Adjuvant or Neo-Adjuvant Therapy | 184 | 192 | 376
  De Novo | 218 | 214 | 432
Independent-Review Facility (IRF)-Determined Disease Status at Screening [Count of Participants; unit: Participants] — A participant was deemed to have measurable disease if they had at least 1 target lesion at screening. Target lesions (maximum of 5 per organ and 10 in total) were selected on the basis of their size (lesions with the longest diameter) and their suitability for accurate repeated measurements (either by imaging techniques or clinically). Any participants with non-target lesions only were deemed to have non-measurable disease. The IRF did not evaluate baseline tumor assessments for any participant without a post-baseline tumor assessment.
  Participants
    Measurable Disease | 343 | 336 | 679
    Non-Measurable Disease | 44 | 43 | 87
    Not Evaluated | 15 | 27 | 42

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Determined by an Independent Review Facility
Description: PFS was defined as the time from randomization to first documented radiographical progressive disease (PD), as determined by an independent review facility (IRF) using RECIST version 1.0, or death from any cause (within 18 weeks of last tumor assessment), whichever occurred first (Kaplan-Meier method). For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum of the LD recorded since treatment started or the appearance of ≥1 new lesion. For non-target lesions, PD was defined as the appearance of ≥1 new lesion or unequivocal progression of existing lesions. Participants without IRF-determined PD or who had not died within 18 weeks of their last IRF-determined, progression-free tumor assessment were censored at the date of the last IRF-reviewed, evaluable tumor assessment; those with no post-baseline tumor assessment and who had not died within 18 weeks of baseline were censored at 1 day.
Time Frame: Tumor assessments every 9 weeks from randomization to IRF-determined PD or death from any cause, whichever occurred first, up to the primary completion date (up to 3 years, 3 months)
Population: Intent-to-Treat (ITT) Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pertuzumab + Trastuzumab + Docetaxel | Placebo + Trastuzumab + Docetaxel
Number analyzed (Participants) | 402 | 406
Months | 18.5 [15 to 23] | 12.4 [10 to 13]
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Docetaxel vs Placebo + Trastuzumab + Docetaxel; The null hypothesis (H0) was that the survival distributions of PFS in the two treatments arms (pertuzumab vs. placebo) are the same. The alternative hypothesis (H1) was that the survival distribution of PFS in the experimental arm (pertuzumab) and control arm (placebo) are different; Test type: Superiority; p < 0.0001, Log Rank (stratified) — Tested at two-sided 5% significance level; Stratified by prior treatment status and region; Cox Proportional Hazard = 0.62, 95% CI 2-sided [0.51 to 0.75] — Hazard ratio is comparing Pertuzumab arm with Placebo arm
Statistical Analysis 2: Comparison: Pertuzumab + Trastuzumab + Docetaxel vs Placebo + Trastuzumab + Docetaxel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Log Rank (unstratified) — Tested at two-sided 5% significance level; Unstratified; Cox Proportional Hazard = 0.63, 95% CI 2-sided [0.52 to 0.76] — Hazard ratio is comparing Pertuzumab arm with Placebo arm

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was the time from randomization to death from any cause, using Kaplan-Meier methodology. Survival data was collected every 18 weeks during the post-treatment follow-up period until death, loss to follow-up, or withdrawal of consent. Those who were alive, lost to follow up, or withdrew consent were censored at the latest date they participated in the study; those without post-baseline data were censored at 1 day. OS analyses were planned to take place at the primary completion date (First Interim), after 385 deaths (Event-Driven Final), and at the end of study (End-of-Study). A second interim OS analysis was planned due to a formal request from the European Medicines Agency. Median [range] time in weeks on study at each OS analysis (Pertuzumab vs. Placebo): First: 77.1 [0.7-165.3] vs. 73.1 [0.4-165.3]; Second: 117.1 [0.7-207.9] vs. 105.9 [0.4-207.9]; Event-Driven Final: 189.9 [0.7-304.1] vs. 140.5 [0.4-301.6]; End-of-Study: 201.8 [0.7-520.0] vs. 138.0 [0.4-514.7].
Time Frame: From randomization to death from any cause, up to each respective analysis data cut-off date (see the Description field for the median time on study per treatment arm)
Population: ITT Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pertuzumab + Trastuzumab + Docetaxel | Placebo + Trastuzumab + Docetaxel
Number analyzed (Participants) | 402 | 406
Months
  End-of-Study OS Analysis | 57.1 [50 to 72] | 40.8 [36 to 48]
  Event-Driven Final OS Analysis | 56.5 [49 to NA] — The upper limit of the 95% CI could not be determined because it was larger than the maximum follow-up time at data cutoff for the analysis. | 40.8 [36 to 48]
  Second Interim OS Analysis | NA [42 to NA] — The median and upper limit of the 95% CI could not be determined because they were larger than the maximum follow-up time at data cutoff for the analysis. | 37.6 [34 to NA] — The upper limit of the 95% CI could not be determined because it was larger than the maximum follow-up time at data cutoff for the analysis.
  First Interim OS Analysis | NA [NA to NA] — The median and lower and upper limits of the 95% CI could not be determined because they were larger than the maximum follow-up time at data cutoff for the analysis. | NA [30 to NA] — The median and upper limit of the 95% CI could not be determined because they were larger than the maximum follow-up time at data cutoff for the analysis.
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Docetaxel vs Placebo + Trastuzumab + Docetaxel; End-of-Study OS Analysis: This end-of-study OS analysis is considered exploratory only as the confirmatory OS analysis for statistical interpretation had previously occurred at the second interim OS analysis; Test type: Superiority — Exploratory; p < 0.0001, Log Rank (stratified) — Exploratory; Stratified by prior treatment status and region; Cox Proportional Hazard = 0.69, 95% CI 2-sided [0.58 to 0.82] — Hazard ratio is comparing Pertuzumab arm with Placebo arm
Statistical Analysis 2: Comparison: Pertuzumab + Trastuzumab + Docetaxel vs Placebo + Trastuzumab + Docetaxel; Event-Driven Final OS Analysis: This final OS analysis was event-driven and planned to take place after a total of 385 deaths had occurred. It is considered exploratory only as the confirmatory OS analysis for statistical interpretation had previously occurred at the second interim OS analysis; Test type: Superiority — Exploratory; p = 0.0002, Log Rank (stratified) — Exploratory; Stratified by prior treatment status and region; Cox Proportional Hazard = 0.68, 95% CI 2-sided [0.56 to 0.84] — Hazard ratio is comparing Pertuzumab arm with Placebo arm
Statistical Analysis 3: Comparison: Pertuzumab + Trastuzumab + Docetaxel vs Placebo + Trastuzumab + Docetaxel; Second Interim OS Analysis: For this second interim OS analysis, the pre-defined O'Brien-Fleming stopping boundary for the Lan-DeMets α-spending function was: HR≤0.739, p≤0.0138; Test type: Superiority; p = 0.0008, Log Rank (stratified) — The threshold for statistical significance was HR≤0.739, p≤0.0138; Stratified by prior treatment status and region; Cox Proportional Hazard = 0.66, 95% CI 2-sided [0.52 to 0.84] — Hazard ratio (HR) is comparing Pertuzumab arm with Placebo arm
Statistical Analysis 4: Comparison: Pertuzumab + Trastuzumab + Docetaxel vs Placebo + Trastuzumab + Docetaxel; First Interim OS Analysis: For this first interim OS analysis, the pre-defined O'Brien-Fleming stopping boundary for the Lan-DeMets α-spending function was: HR≤0.603, p≤0.0012; Test type: Superiority; p = 0.0050, Log Rank (stratified) — The threshold for statistical significance was HR≤0.603, p≤0.0012; Stratified by prior treatment status and region; Cox Proportional Hazard = 0.64, 95% CI 2-sided [0.47 to 0.88] — Hazard ratio (HR) is comparing pertuzumab with placebo arms

3. Secondary Outcome: Progression-Free Survival (PFS) Determined by the Investigator
Description: PFS was defined as the time from randomization to first documented radiographical progressive disease (PD), as determined by the investigator using RECIST version 1.0, or death from any cause (within 18 weeks of last tumor assessment), whichever occurred first (Kaplan-Meier method). For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum of the LD recorded since treatment started or the appearance of ≥1 new lesion. For non-target lesions, PD was defined as the appearance of ≥1 new lesion or unequivocal progression of existing lesions. Participants without PD or who had not died within 18 weeks of their last investigator-determined, progression-free tumor assessment were censored at the date of the last investigator tumor assessment; those with no post-baseline tumor assessment and who had not died within 18 weeks of baseline were censored at 1 day.
Time Frame: Tumor assessments every 9 weeks from randomization to investigator-determined PD or death from any cause, whichever occurred first (median [range] time on study in pertuzumab vs. placebo arms: 201.8 [0.7-520.0] weeks vs. 138.0 [0.4-514.7] weeks)
Population: Intent-to-treat population: All randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pertuzumab + Trastuzumab + Docetaxel | Placebo + Trastuzumab + Docetaxel
Number analyzed (Participants) | 402 | 406
Months | 18.7 [17 to 22] | 12.4 [10 to 14]
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Docetaxel vs Placebo + Trastuzumab + Docetaxel; PFS by Investigator - Stratified; Test type: Superiority; p < 0.0001, Log Rank (stratified); Stratified by prior treatment status and region; Cox Proportional Hazard = 0.69, 95% CI 2-sided [0.59 to 0.81] — Hazard ratio is comparing Pertuzumab arm with Placebo arm

4. Secondary Outcome: Objective Response Determined by an Independent Review Facility
Description: An objective response was defined as the percentage of participants with confirmed best overall response of complete response (CR) or partial response (PR) determined by an independent review facility (IRF) using RECIST v1.0 on two consecutive occasions ≥4 weeks apart. For target lesions, CR: disappearance of all target lesions; PR: ≥30% decrease in the sum of the longest diameter (LD) of target lesions (baseline sum LD as reference); PD: ≥20% increase in the sum of the LD of target lesions (smallest sum of the LD recorded as reference) or appearance of ≥1 new lesion; SD: neither sufficient shrinkage to qualify for PR nor sufficient increase for PD. For non-target lesions, CR: disappearance of all non-target lesions; Incomplete/SD: persistence of ≥1 non-target lesions; PD: unequivocal progression of existing non-target lesions. 95% confidence intervals (CI) were calculated only for clinical responses using the Pearson-Clopper method.
Time Frame: Tumor assessments every 9 weeks from Baseline until IRF-determined progressive disease (PD), death, or first administration of next line of anti-cancer therapy (whichever occurred first), up to the primary completion date (up to 3 years, 3 months)
Population: ITT Population: All randomized participants; only participants with IRF-determined measurable disease at baseline (i.e., ≥1 target lesion) were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Pertuzumab + Trastuzumab + Docetaxel | Placebo + Trastuzumab + Docetaxel
Number analyzed (Participants) | 343 | 336
Percentage of patients
  Objective Response (CR + PR) | 80.2 [75.6 to 84.3] | 69.3 [64.1 to 74.2]
  Complete Response (CR) | 5.5 [3.4 to 8.5] | 4.2 [2.3 to 6.9]
  Partial Response (PR) | 74.6 [69.7 to 79.2] | 65.2 [59.8 to 70.3]
  Stable Disease (SD) | 14.6 [11.0 to 18.8] | 20.8 [16.6 to 25.6]
  Progressive Disease (PD) | 3.8 [2.0 to 6.4] | 8.3 [5.6 to 11.8]
  Unable to Assess (UA) | 0.6 [0.1 to 2.1] | 0.6 [0.1 to 2.1]
  Missing (No Assessment) | 0.9 [NA to NA] — 95% confidence intervals were calculated only for clinical responses. | 0.9 [NA to NA] — 95% confidence intervals were calculated only for clinical responses.
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Docetaxel vs Placebo + Trastuzumab + Docetaxel; Difference in Objective Response (CR + PR) Between Arms; Test type: Superiority; p = 0.0011, Mantel Haenszel; Stratified by prior treatment status and region; Difference in Objective Response Rates = 10.83, 95% CI 2-sided [4.2 to 17.5] — Difference in the objective response rates between arms is calculated as Pertuzumab arm minus Placebo arm. The 95% CI was calculated using the Hauck-Anderson method
Statistical Analysis 2: Comparison: Pertuzumab + Trastuzumab + Docetaxel vs Placebo + Trastuzumab + Docetaxel; Odds Ratio for Objective Response (CR + PR); Test type: Superiority; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.26 to 2.54]

5. Secondary Outcome: Duration of Objective Response Determined by an Independent Review Facility
Description: Duration of objective response (estimated using the Kaplan-Meier method) was defined as the time from the initial confirmed complete response (CR) or partial response (PR), the date of tumor assessment at which the CR/PR was first detected by the independent review facility (IRF) using RECIST version 1.0, until the date of IRF-determined progressive disease (PD), death from any cause within 18 weeks of the last tumor assessment, or first administration of next line of anti-cancer therapy (whichever occurred first). If the visit when the initial CR or PR was observed spanned multiple dates, the latest date was used. Only participants in the ITT analysis population with an IRF-determined objective response (CR or PR), observed prior to IRF-assessed PD, death or next line of anti-cancer therapy, were included in the analysis. Participants who did not progress or die after they had a confirmed response were censored at the date of their last IRF-evaluable tumor measurement.
Time Frame: From initial IRF-confirmed objective response until IRF-determined progressive disease (PD), death, or first administration of next line of anti-cancer therapy (whichever occurred first), up to the primary completion date (up to 3 years, 3 months)
Population: ITT Population: All randomized participants; only participants with IRF-determined measurable disease at baseline (i.e., ≥1 target lesion) that had an objective response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pertuzumab + Trastuzumab + Docetaxel | Placebo + Trastuzumab + Docetaxel
Number analyzed (Participants) | 275 | 233
Weeks | 87.6 [71 to 106] | 54.1 [46 to 64]
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Docetaxel vs Placebo + Trastuzumab + Docetaxel; Test type: Superiority; Cox Proportional Hazard = 0.66, 95% CI 2-sided [0.51 to 0.85]

6. Secondary Outcome: Time to Symptom Progression
Description: Time to symptom progression was defined as the time from randomization to the first symptom progression as measured by the Functional Assessment of Cancer Therapy-for patients with Breast Cancer (FACT-B) questionnaire with the Trial Outcomes Index-Physical/Functional/Breast (TOI-PFB) subscale. The FACT-B TOI-PFB subscale contains 24 items from 3 subsections of the FACT-B questionnaire: Physical well-being, functional well-being, and additional concerns for breast cancer patients (breast cancer subscale [BCS]). All items in the questionnaire were rated by the patient on a 5-point scale ranging from 0 ("not at all") to 4 ("very much"). The total score ranged from 0 to 96. A higher score indicates better perceived quality of life. A positive change score from baseline indicates improvement. Symptom progression was defined as a decrease from baseline of 5 points or more.
Time Frame: Every 9 weeks from Baseline until investigator-determined progressive disease, up to the primary completion date (up to 3 years, 3 months)
Population: ITT population: All randomized participants; only female participants were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pertuzumab + Trastuzumab + Docetaxel | Placebo + Trastuzumab + Docetaxel
Number analyzed (Participants) | 402 | 404
Weeks | 18.4 [18 to 27] | 18.3 [18 to 27]
Statistical Analysis 1: Comparison: Pertuzumab + Trastuzumab + Docetaxel vs Placebo + Trastuzumab + Docetaxel; Test type: Superiority; p = 0.7161, Log Rank (stratified) — Stratified by prior treatment status and region; Cox Proportional Hazard = 0.97, 95% CI 2-sided [0.81 to 1.16] — Hazard ratio is comparing Pertuzumab arm with Placebo arm

7. Secondary Outcome: Overall Number of Participants Who Experienced at Least One Adverse Event, Including Serious and Non-Serious Adverse Events, by Most Severe Intensity (According to NCI-CTCAE v3.0) During the Treatment Period
Description: Adverse event (AE) severity was assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 3.0 (NCI-CTCAE v3.0); if the AE was not specifically listed, the following grades of severity were used: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening or disabling; and Grade 5 = death. Severe and serious are not synonymous. Severity refers to the intensity of an AE, whereas a serious AE must meet criteria set out in the protocol; both were independently assessed for each AE. Only the most severe intensity was counted for multiple occurrences of the same AE in one participant. AEs reported prior to first crossover treatment were included in the Placebo arm, and in the Crossover arm after that date, for participants who crossed over from placebo to pertuzumab. Median [range] time on study treatment per arm: Placebo: 49.3 [0.3-514.7] weeks; Pertuzumab: 75.7 [0.6-519.6] weeks; Crossover: 129.9 [0.3-322.3] weeks.
Time Frame: Placebo arm: Baseline to last dose of study treatment +42 days (or crossover date); Pertuzumab arm: Baseline to last dose of study treatment +42 days; Crossover arm: Crossover date to last dose of study treatment +42 days (see Description - time per arm)
Population: Safety Population: All participants who received at least one dose of any study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo + Trastuzumab + Docetaxel: This is the placebo safety population, which includes participants who received study treatment with placebo at every cycle. Participants received placebo IV q3w and trastuzumab 6 mg/kg IV q3w, plus docetaxel 75 mg/m^2 IV q3w (for at least 6 cycles; 1 cycle was 21 days). After Cycle 6, continuation of docetaxel treatment was at the discretion of the participant and treating physician. Participants remained in the treatment phase of the study until investigator-assessed radiographic or clinical evidence of disease progression, unmanageable toxicity, or study termination and were followed for survival until death, loss to follow-up, withdrawal of consent, or study termination.
- Pertuzumab + Trastuzumab + Docetaxel: This is the pertuzumab safety population, which includes participants who received at least one dose of study treatment with pertuzumab. Participants received pertuzumab 420 milligrams (mg) intravenously (IV) once every 3 weeks (q3w) and trastuzumab 6 milligrams per kilogram (mg/kg) IV q3w, plus docetaxel 75 milligrams per square metre of body surface (mg/m^2) IV q3w (for at least 6 cycles; 1 cycle was 21 days). After Cycle 6, continuation of docetaxel treatment was at the discretion of the participant and treating physician. Participants remained in the treatment phase of the study until investigator-assessed radiographic or clinical evidence of disease progression, unmanageable toxicity, or study termination and were followed for survival until death, loss to follow-up, withdrawal of consent, or study termination.
- Crossover From Placebo to Pertuzumab: Fifty of 406 participants (12.3%) randomized to the placebo treatment arm whose disease had not progressed crossed over to an open-label pertuzumab treatment group between July 2012 and November 2018. Participants received pertuzumab administered as an IV loading dose of 840 mg at cycle 1 then 420 mg IV every q3w. Trastuzumab and docetaxel doses continued in accordance with the pre-crossover placebo treatment regimens and according to dosing specifications indicated in the study protocol. Participants remained in the treatment phase of the study until investigator-assessed radiographic or clinical evidence of disease progression, unmanageable toxicity, or study termination and were followed for survival until death, loss to follow-up, withdrawal of consent, or study termination.
Arm/Group | Placebo + Trastuzumab + Docetaxel | Pertuzumab + Trastuzumab + Docetaxel | Crossover From Placebo to Pertuzumab
Number analyzed (Participants) | 396 | 408 | 50
Participants
  At Least One Serious AE - All Grades | 116 | 160 | 10
  At Least One Non-Serious AE - All Grades | 386 | 400 | 45
  At Least One AE - All Grades | 391 | 408 | 47
  At Least One AE - Grade 1 | 368 | 386 | 44
  At Least One AE - Grade 2 | 350 | 383 | 34
  At Least One AE - Grade 3 | 229 | 264 | 11
  At Least One AE - Grade 4 | 158 | 167 | 1
  At Least One AE - Grade 5 | 12 | 8 | 1

8. Secondary Outcome: Overall Number of Adverse Events by Severity (NCI-CTCAE v3.0 All Grades and Grades 3 to 5) Per 100 Patient-Years of Exposure During the Treatment Period
Description: Adverse event (AE) severity, including serious and non-serious AEs, was assessed according to the NCI-CTCAE version 3.0; if the AE was not specifically listed, the following grades of severity were used: Grade 1 is mild; Grade 2 is moderate; Grade 3 is severe; Grade 4 is life-threatening or disabling; and Grade 5 is death. Multiple occurrences of the same AE in 1 participant were counted multiple times. Only AEs that started during the overall study treatment period were included. The cutoff date for inclusion of events and for calculation of patient-years was the date of the most recent follow-up of the participant, defined as the last available date during the treatment period, excluding pre-treatment and safety follow-up data. Confidence intervals were calculated assuming the number of events followed a Poisson distribution. Data reported prior to the date of first crossover treatment were included under the Placebo arm for participants who crossed over from placebo to pertuzumab.
Time Frame: From Baseline to 42 days after the last dose of study treatment (total patient-years of exposure on study treatment in Placebo vs. Pertuzumab arms: 526.81 vs. 989.88 patient-years)
Population: Safety Population: All participants who received at least one dose of any study medication.
Measure: Number (90% Confidence Interval); unit: Events per 100 patient-years
Units Other Than Participants: Adverse Events
Groups:
- Placebo + Trastuzumab + Docetaxel: This is the placebo safety population, which includes participants who received study treatment with placebo at every cycle. Participants received placebo IV q3w and trastuzumab 6 mg/kg IV q3This is the placebo safety population, which includes participants who received study treatment with placebo at every cycle. Participants received placebo IV q3w and trastuzumab 6 mg/kg IV q3w, plus docetaxel 75 mg/m^2 IV q3w (for at least 6 cycles; 1 cycle was 21 days). After Cycle 6, continuation of docetaxel treatment was at the discretion of the participant and treating physician. Participants remained in the treatment phase of the study until investigator-assessed radiographic or clinical evidence of disease progression, unmanageable toxicity, or study termination and were followed for survival until death, loss to follow-up, withdrawal of consent, or study termination.
Arm/Group | Placebo + Trastuzumab + Docetaxel | Pertuzumab + Trastuzumab + Docetaxel
Number analyzed (Participants) | 396 | 408
Number analyzed (Adverse Events) | 9062 | 11908
Events per 100 patient-years
  All Grades | 1720.2 [1690.6 to 1750.2] | 1203.0 [1184.9 to 1221.3]
  Grades 3 to 5: number analyzed (Adverse Events) | 1187 | 1304
  Grades 3 to 5 | 225.3 [214.7 to 236.4] | 131.7 [125.8 to 137.9]

9. Secondary Outcome: Cardiac-Related AEs to Monitor: Number of Participants Who Experienced at Least One Symptomatic Left Ventricular Dysfunction (LVD), Any LVD, or Serious AE Suggestive of Congestive Heart Failure by Severity During the Treatment Period
Description: Cardiac-related adverse events (AEs) to monitor during the study included investigator-assessed symptomatic left ventricular dysfunction (LVD), any LVD, or a serious adverse event (SAE) suggestive of congestive heart failure (CHF). All cardiac-related AEs were graded for severity according to NCI-CTCAE v3.0. Asymptomatic (Grades 1-2) and symptomatic (Grades 3-5) left ventricular systolic dysfunction (LVSD) both coded to the MedDRA preferred term LVD. Investigator-assessed events of symptomatic LVD were also graded for severity of symptoms according to Classes I (least severe) to IV (most severe) of the New York Heart Association (NYHA) Classification. SAEs suggestive of CHF were identified as serious events from the Standardized MedDRA Query (SMQ) (Wide) 'Cardiac Failure'. Median [range] time on study treatment per arm: Placebo: 49.3 [0.3-514.7] weeks; Pertuzumab: 75.7 [0.6-519.6] weeks; Crossover: 129.9 [0.3-322.3] weeks.
Time Frame: as for outcome 7
Population: Safety Population: All participants who received at least one dose of any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Trastuzumab + Docetaxel | Pertuzumab + Trastuzumab + Docetaxel | Crossover From Placebo to Pertuzumab
Number analyzed (Participants) | 396 | 408 | 50
Participants
  Symptomatic LVD(Investigator)-All NYHA Classes | 7 | 6 | 1
  Symptomatic LVD(Investigator)-NYHA Classes III/IV | 4 | 4 | 1
  Any LVD - All NCI-CTCAE Grades | 34 | 32 | 3
  Any LVD - NCI-CTCAE Grade ≥3 | 13 | 6 | 2
  SAE Suggestive of CHF - All NCI-CTCAE Grades | 8 | 8 | 1
  SAE Suggestive of CHF - NCI-CTCAE Grade ≥3 | 7 | 7 | 1

10. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event to Monitor (Excluding Cardiac-Related AEs) by Severity During the Treatment Period
Description: The clinical diagnoses listed in this table, excluding cardiac safety (summarized separately), were also selected as adverse events (AEs) to monitor based on clinical and nonclinical data for pertuzumab and the safety profile established for trastuzumab, monoclonal antibodies in general, and potential effects associated with HER receptor inhibition. Search strategies were defined by single or aggregate MedDRA Preferred Terms (PT) through Standardized MedDRA Queries (SMQ), where possible, or based on Roche AE Group Terms (AEGT). Diarrhoea AEs: High-Level Term (HLT) 'Diarrhoea (excl. infective)' and PT 'Diarrhoea infectious'. Leukopenic and Febrile Neutropenic Infections: AEs from 'Infections & Infestations' with start ≤14 days after start date of Grade ≥3 AEs in SMQ(narrow) 'Leukopenia' or PT 'Febrile neutropenia', respectively. Median [range] time on study treatment per arm: Placebo: 49.3 [0.3-514.7] weeks; Pertuzumab: 75.7 [0.6-519.6] weeks; Crossover: 129.9 [0.3-322.3] weeks.
Time Frame: as for outcome 7
Population: Safety Population: All participants who received at least one dose of any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Trastuzumab + Docetaxel | Pertuzumab + Trastuzumab + Docetaxel | Crossover From Placebo to Pertuzumab
Number analyzed (Participants) | 396 | 408 | 50
Participants
  Diarrhoea (HLT+PT) - All Grades | 191 | 280 | 25
  Diarrhoea (HLT+PT) - Grade ≥3 | 20 | 40 | 1
  Rash (AEGT) - All Grades | 155 | 213 | 18
  Rash (AEGT) - Grade ≥3 | 6 | 15 | 0
  Leukopenia (SMQ-narrow) - All Grades | 231 | 257 | 1
  Leukopenia (SMQ-narrow) - Grade ≥3 | 211 | 238 | 0
  Leukopenic Infection (PTs) - All Grades | 38 | 53 | 0
  Leukopenic Infection (PTs) - Grade ≥3 | 9 | 18 | 0
  Febrile Neutropenic Infection (PTs) - All Grades | 3 | 14 | 0
  Febrile Neutropenic Infection (PTs) - Grade ≥3 | 1 | 6 | 0
  Anaphylaxis and Hypersensitivity (AEGT)-All Grades | 37 | 48 | 1
  Anaphylaxis and Hypersensitivity (AEGT)-Grade ≥3 | 10 | 9 | 0
  Interstitial Lung Disease (SMQ-narrow) -All Grades | 6 | 10 | 1
  Interstitial Lung Disease (SMQ-narrow) -Grade ≥3 | 2 | 3 | 0
  QT Prolongation (SMQ-wide) - All Grades | 5 | 16 | 0
  QT Prolongation (SMQ-wide) - Grade ≥3 | 1 | 7 | 0
  Mucositis (AEGT) - All Grades | 154 | 208 | 12
  Mucositis (AEGT) - Grade ≥3 | 8 | 14 | 0
  Drug-Related Hepatic Disorder(SMQ-wide)-All Grades | 43 | 47 | 0
  Drug-Related Hepatic Disorder (SMQ-wide)-Grade ≥3 | 5 | 8 | 0

11. Secondary Outcome: Overall Number of Participants Who Experienced at Least One Adverse Event Leading to Discontinuation of Any or All Study Medication
Description: Participants could continue study treatment with pertuzumab/placebo plus trastuzumab when docetaxel was discontinued due to an adverse event (AE). Discontinuation of pertuzumab/placebo or trastuzumab due to an AE led to discontinuation of all study medication. The number of participants who discontinued any study medication due to an AE includes those who discontinued all study medication and those who discontinued docetaxel only and then continued on targeted therapy (note: some of these participants may have subsequently discontinued all treatment due to a separate AE). Multiple occurrences of the same adverse event in 1 participant was counted only once. AEs reported prior to first crossover treatment were included in the Placebo arm, and after that date in the Crossover arm, for those who crossed over from placebo to pertuzumab. Median [range] time on study treatment per arm: Placebo: 49.3 [0.3-514.7] weeks; Pertuzumab: 75.7 [0.6-519.6] weeks; Crossover: 129.9 [0.3-322.3] weeks.
Time Frame: as for outcome 7
Population: Safety Population: All participants who received at least one dose of any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Trastuzumab + Docetaxel | Pertuzumab + Trastuzumab + Docetaxel | Crossover From Placebo to Pertuzumab
Number analyzed (Participants) | 396 | 408 | 50
Participants
  AE Leading to Discontinuation-Any Study Medication | 114 | 131 | 5
  AE Leading to Discontinuation-All Study Medication | 24 | 39 | 4

12. Secondary Outcome: Overall Number of Participants Who Experienced at Least One Adverse Event That Resulted in Interruption or Modification of Any Study Medication
Description: Pertuzumab, trastuzumab, and docetaxel administration could have been delayed to assess or treat adverse events (AEs). Docetaxel dose reduction was allowed for myelosuppression, hepatic dysfunction, and other toxicities. No dose reduction was allowed for pertuzumab or trastuzumab. Multiple occurrences of the same adverse event in one participant was counted only once. AEs reported prior to first crossover treatment were included in the Placebo arm, and after that date in the Crossover arm, for participants who crossed over from placebo to pertuzumab. Median [range] time on study treatment per arm: Placebo: 49.3 [0.3-514.7] weeks; Pertuzumab: 75.7 [0.6-519.6] weeks; Crossover: 129.9 [0.3-322.3] weeks
Time Frame: as for outcome 7
Population: Safety Population: All participants who received at least one dose of any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Trastuzumab + Docetaxel | Pertuzumab + Trastuzumab + Docetaxel | Crossover From Placebo to Pertuzumab
Number analyzed (Participants) | 396 | 408 | 50
Participants | 217 | 265 | 16

13. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event During the Post-Treatment Follow-Up Period
Description: The post-treatment period was defined as the period following the treatment discontinuation visit. Only the following new adverse events (AEs) should have been reported during the post-treatment follow-up period: 1. Cardiac events (regardless of causality or seriousness) that started up to 1 year after the last dose, except for symptomatic left ventricular systolic dysfunction (regardless of causality) that started up to 3 years after the last dose; and 2. Treatment-related serious AEs, regardless of start date. AEs are listed by Medical Dictionary for Regulatory Activities, Version 21.1 (MedDRA v21.1) System Organ Class (SOC) and Preferred Term (PT); PTs fall under the SOC that is listed immediately above it in the table. Multiple occurrences of the same AE in one participant was counted only once. AEs reported prior to first crossover treatment were included in the Placebo arm, and after that date in the Crossover arm, for participants who crossed over from placebo to pertuzumab.
Time Frame: From Day 43 after discontinuation of all study medication to end of post-treatment follow-up period (up to 3 years)
Population: Safety Population: All participants who received at least one dose of any study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Trastuzumab + Docetaxel | Pertuzumab + Trastuzumab + Docetaxel | Crossover From Placebo to Pertuzumab
Number analyzed (Participants) | 396 | 408 | 50
Participants
  Total with at Least One AE During Post-Treatment | 18 | 17 | 3
  Cardiac Disorders (SOC) | 8 | 9 | 1
  Left Ventricular Dysfunction (PT) | 6 | 5 | 1
  Cardiac Failure (PT) | 0 | 2 | 0
  Bundle Branch Block Left (PT) | 0 | 1 | 0
  Cardiopulmonary Failure (PT) | 1 | 0 | 0
  Myocardial Ischaemia (PT) | 1 | 0 | 0
  Pericardial Effusion (PT) | 0 | 1 | 0
  Prinzmetal Angina (PT) | 1 | 0 | 0
  General Disorders & Admin. Site Conditions (SOC) | 3 | 2 | 0
  Oedema Peripheral (PT) | 2 | 1 | 0
  Asthenia (PT) | 1 | 0 | 0
  Influenza Like Illness (PT) | 0 | 1 | 0
  Infections & Infestations (SOC) | 0 | 0 | 2
  Influenza (PT) | 0 | 0 | 1
  Viral Infection (PT) | 0 | 0 | 1
  Abscess Limb (PT) | 0 | 1 | 0
  Nasopharyngitis (PT) | 1 | 0 | 0
  Subcutaneous Abscess (PT) | 0 | 1 | 0
  Musculoskeletal & Connective Tissue Disorders(SOC) | 0 | 0 | 1
  Back Pain (PT) | 0 | 0 | 1
  Pain in Extremity (PT) | 1 | 0 | 0
  Nervous System Disorders (SOC) | 2 | 2 | 0
  Neuropathy Peripheral (PT) | 1 | 1 | 0
  Cognitive Disorder (PT) | 1 | 0 | 0
  Dizziness (PT) | 0 | 1 | 0
  Headache (PT) | 0 | 1 | 0
  Respiratory, Thoracic & Mediastinal Disorders(SOC) | 2 | 1 | 0
  Cough (PT) | 1 | 0 | 0
  Dyspnoea (PT) | 1 | 0 | 0
  Rhinitis Allergic (PT) | 0 | 1 | 0
  Skin & Subcutaneous Tissue Disorders (SOC) | 1 | 2 | 0
  Erythema (PT) | 0 | 1 | 0
  Nail Disorder (PT) | 1 | 0 | 0
  Rash Macular (PT) | 0 | 1 | 0
  Blood & Lymphatic System Disorders (SOC) | 1 | 1 | 0
  Febrile Neutropenia (PT) | 1 | 0 | 0
  Leukopenia (PT) | 0 | 1 | 0
  Gastrointestinal Disorders (SOC) | 0 | 2 | 0
  Diarrhoea (PT) | 0 | 1 | 0
  Stomatitis (PT) | 0 | 1 | 0
  Endocrine Disorders (SOC) | 1 | 0 | 0
  Thyroid Mass (PT) | 1 | 0 | 0
  Eye Disorders (SOC) | 1 | 0 | 0
  Retinal Detachment (PT) | 1 | 0 | 0
  Immune System Disorders (SOC) | 0 | 1 | 0
  Iodine Allergy (PT) | 0 | 1 | 0
  Investigations (SOC) | 1 | 0 | 0
  Aspartate Aminotransferase Increased (PT) | 1 | 0 | 0
  Renal & Urinary Disorders (SOC) | 0 | 1 | 0
  Dysuria (PT) | 0 | 1 | 0
  Reproductive System & Breast Disorders (SOC) | 0 | 1 | 0
  Breast Induration (PT) | 0 | 1 | 0
  Vascular Disorders (SOC) | 0 | 1 | 0
  Venous Thrombosis (PT) | 0 | 1 | 0

14. Secondary Outcome: Number of Participants by Categories for the Maximum Absolute Decrease From Baseline in LVEF Value During the Treatment Period
Description: All participants were required to have an left ventricular ejection fraction (LVEF) ≥50% at baseline, as measured by echocardiogram (preferred) or multiple-gated acquisition (MUGA) scan. The same method of LVEF assessment and the same institution/facility used at baseline was used throughout the study, to the extent possible. The baseline value was defined as the last valid value recorded during the pre-treatment period before or on study Day 1. The maximum absolute decrease in LVEF value was defined as the lowest post-baseline value up to the end of the overall study treatment period. Data reported prior to first crossover treatment were included in the Placebo arm, and after that date in the Crossover arm, for participants who crossed over from placebo to pertuzumab. Median [range] time on study treatment per arm: Placebo: 49.3 [0.3-514.7] weeks; Pertuzumab: 75.7 [0.6-519.6] weeks; Crossover: 129.9 [0.3-322.3] weeks.
Time Frame: Every 9 weeks from the date of randomization until Treatment Discontinuation Visit (see Description for time on study treatment per arm)
Population: Safety Population: All participants who received at least one dose of any study medication. Only participants with evaluable LVEF assessments during the overall study treatment period were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Trastuzumab + Docetaxel | Pertuzumab + Trastuzumab + Docetaxel | Crossover From Placebo to Pertuzumab
Number analyzed (Participants) | 396 | 408 | 50
Participants
  LVEF Increase/No Change/Decrease FromBL <10%Points: number analyzed (Participants) | 378 | 394 | 49
  LVEF Increase/No Change/Decrease FromBL <10%Points | 252 | 249 | 30
  LVEF <50% and Decrease From BL ≥10% to <15% Points: number analyzed (Participants) | 378 | 394 | 49
  LVEF <50% and Decrease From BL ≥10% to <15% Points | 9 | 7 | 0
  LVEF <50% and Decrease From BL ≥15% Points: number analyzed (Participants) | 378 | 394 | 49
  LVEF <50% and Decrease From BL ≥15% Points | 19 | 21 | 3
  LVEF ≥50% and Decrease From BL ≥10% Points: number analyzed (Participants) | 378 | 394 | 49
  LVEF ≥50% and Decrease From BL ≥10% Points | 95 | 115 | 15
  No Baseline (BL) LVEF Value: number analyzed (Participants) | 378 | 394 | 49
  No Baseline (BL) LVEF Value | 3 | 2 | 1

15. Secondary Outcome: Baseline LVEF Value and Change in LVEF From Baseline at Maximum Absolute Decrease Value During the Treatment Period
Description: All participants were required to have a left ventricular ejection fraction (LVEF) ≥50% at baseline, as measured by echocardiogram (preferred) or multiple-gated acquisition (MUGA) scan. The same method of LVEF assessment and the same institution/facility used at baseline was used throughout the study, to the extent possible. The baseline value was defined as the last valid value recorded during the pre-treatment period before or on study Day 1. The maximum absolute decrease in LVEF value was defined as the lowest post-baseline value up to the end of the overall study treatment period. Only data reported prior to the date of first crossover treatment were included for participants who crossed over from placebo to pertuzumab.
Time Frame: Every 9 weeks from the date of randomization until Treatment Discontinuation Visit (median [range] time on study treatment per arm: Placebo: 49.3 [0.3-514.7] weeks; Pertuzumab: 75.7 [0.6-519.6] weeks)
Population: Safety Population: All participants who received at least one dose of any study medication. Only participants with evaluable LVEF assessments at baseline (BL) or at BL and post-BL (for change in LVEF from BL at max. decrease) were included in the analyses.
Measure: Mean (Standard Deviation); unit: Percentage points of LVEF
Arm/Group | Placebo + Trastuzumab + Docetaxel | Pertuzumab + Trastuzumab + Docetaxel
Number analyzed (Participants) | 396 | 408
Percentage points of LVEF
  Baseline (BL) LVEF Value: number analyzed (Participants) | 393 | 406
  Baseline (BL) LVEF Value | 65.6 (6.51) | 64.8 (6.71)
  Change in LVEF From BL at Maximum Decrease Value: number analyzed (Participants) | 375 | 392
  Change in LVEF From BL at Maximum Decrease Value | -7.3 (7.15) | -7.5 (7.75)
Statistical Analysis 1: Comparison: Placebo + Trastuzumab + Docetaxel vs Pertuzumab + Trastuzumab + Docetaxel; Wilcoxon Test of Maximum Decrease in LVEF From BL; Test type: Other; p = 0.7174, Wilcoxon Rank Sum Test

16. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Blood Biochemistry Tests by Highest Grade According to NCI-CTCAE v3.0 During the Treatment Period
Description: Clinical laboratory tests for blood biochemistry parameters were performed at local laboratories; any abnormal values (High or Low) were based on local laboratory normal ranges. Laboratory abnormalities are presented by the highest grade according to NCI-CTCAE v3.0. Not every abnormal laboratory value qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy. Median [range] time on study treatment per arm: Placebo: 49.3 [0.3-514.7] weeks; Pertuzumab: 75.7 [0.6-519.6] weeks; Crossover: 129.9 [0.3-322.3] weeks. ALP = alkaline phosphatase; GGT = gamma-glutamyl transferase; SGOT = serum glutamic-oxaloacetic transaminase; SGPT = serum glutamic-pyruvic transaminase
Time Frame: On Day 1 of every treatment cycle (1 cycle is 21 days) until Treatment Discontinuation Visit (see Description for time on study treatment per arm)
Population: Safety Population: All participants who received at least one dose of any study medication. Only participants with at least one valid laboratory value for any given parameter during the overall study treatment period were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Trastuzumab + Docetaxel | Pertuzumab + Trastuzumab + Docetaxel | Crossover From Placebo to Pertuzumab
Number analyzed (Participants) | 396 | 408 | 50
Participants
  Albumin (g/L) - Low, Any Grade (Gr.): number analyzed (Participants) | 385 | 396 | 49
  Albumin (g/L) - Low, Any Grade (Gr.) | 163 | 196 | 15
  Albumin (g/L) - Low, Gr. 1: number analyzed (Participants) | 385 | 396 | 49
  Albumin (g/L) - Low, Gr. 1 | 113 | 132 | 10
  Albumin (g/L) - Low, Gr. 2: number analyzed (Participants) | 385 | 396 | 49
  Albumin (g/L) - Low, Gr. 2 | 46 | 58 | 4
  Albumin (g/L) - Low, Gr. 3: number analyzed (Participants) | 385 | 396 | 49
  Albumin (g/L) - Low, Gr. 3 | 4 | 6 | 1
  Albumin (g/L) - Low, Gr. 4: number analyzed (Participants) | 385 | 396 | 49
  Albumin (g/L) - Low, Gr. 4 | 0 | 0 | 0
  ALP (U/L) - High, Any Gr.: number analyzed (Participants) | 388 | 400 | 49
  ALP (U/L) - High, Any Gr. | 184 | 210 | 17
  ALP (U/L) - High, Gr. 1: number analyzed (Participants) | 388 | 400 | 49
  ALP (U/L) - High, Gr. 1 | 158 | 177 | 17
  ALP (U/L) - High, Gr. 2: number analyzed (Participants) | 388 | 400 | 49
  ALP (U/L) - High, Gr. 2 | 19 | 24 | 0
  ALP (U/L) - High, Gr. 3: number analyzed (Participants) | 388 | 400 | 49
  ALP (U/L) - High, Gr. 3 | 7 | 9 | 0
  ALP (U/L) - High, Gr. 4: number analyzed (Participants) | 388 | 400 | 49
  ALP (U/L) - High, Gr. 4 | 0 | 0 | 0
  Calcium (mmol/L) - Low, Any Gr.: number analyzed (Participants) | 387 | 399 | 49
  Calcium (mmol/L) - Low, Any Gr. | 156 | 203 | 14
  Calcium (mmol/L) - Low, Gr. 1: number analyzed (Participants) | 387 | 399 | 49
  Calcium (mmol/L) - Low, Gr. 1 | 107 | 139 | 11
  Calcium (mmol/L) - Low, Gr. 2: number analyzed (Participants) | 387 | 399 | 49
  Calcium (mmol/L) - Low, Gr. 2 | 45 | 49 | 0
  Calcium (mmol/L) - Low, Gr. 3: number analyzed (Participants) | 387 | 399 | 49
  Calcium (mmol/L) - Low, Gr. 3 | 3 | 7 | 1
  Calcium (mmol/L) - Low, Gr. 4: number analyzed (Participants) | 387 | 399 | 49
  Calcium (mmol/L) - Low, Gr. 4 | 1 | 8 | 2
  Calcium (mmol/L) - High, Any Gr.: number analyzed (Participants) | 387 | 399 | 49
  Calcium (mmol/L) - High, Any Gr. | 54 | 79 | 12
  Calcium (mmol/L) - High, Gr. 1: number analyzed (Participants) | 387 | 399 | 49
  Calcium (mmol/L) - High, Gr. 1 | 50 | 65 | 7
  Calcium (mmol/L) - High, Gr. 2: number analyzed (Participants) | 387 | 399 | 49
  Calcium (mmol/L) - High, Gr. 2 | 0 | 2 | 1
  Calcium (mmol/L) - High, Gr. 3: number analyzed (Participants) | 387 | 399 | 49
  Calcium (mmol/L) - High, Gr. 3 | 3 | 2 | 0
  Calcium (mmol/L) - High, Gr. 4: number analyzed (Participants) | 387 | 399 | 49
  Calcium (mmol/L) - High, Gr. 4 | 1 | 10 | 4
  Creatinine (umol/L) - High, Any Gr.: number analyzed (Participants) | 390 | 402 | 49
  Creatinine (umol/L) - High, Any Gr. | 317 | 346 | 38
  Creatinine (umol/L) - High, Gr. 1: number analyzed (Participants) | 390 | 402 | 49
  Creatinine (umol/L) - High, Gr. 1 | 271 | 279 | 27
  Creatinine (umol/L) - High, Gr. 2: number analyzed (Participants) | 390 | 402 | 49
  Creatinine (umol/L) - High, Gr. 2 | 44 | 54 | 9
  Creatinine (umol/L) - High, Gr. 3: number analyzed (Participants) | 390 | 402 | 49
  Creatinine (umol/L) - High, Gr. 3 | 2 | 6 | 0
  Creatinine (umol/L) - High, Gr. 4: number analyzed (Participants) | 390 | 402 | 49
  Creatinine (umol/L) - High, Gr. 4 | 0 | 7 | 2
  Fasting Glucose (mmol/L) - Low, Any Gr.: number analyzed (Participants) | 387 | 400 | 49
  Fasting Glucose (mmol/L) - Low, Any Gr. | 42 | 75 | 6
  Fasting Glucose (mmol/L) - Low, Gr. 1: number analyzed (Participants) | 387 | 400 | 49
  Fasting Glucose (mmol/L) - Low, Gr. 1 | 32 | 61 | 4
  Fasting Glucose (mmol/L) - Low, Gr. 2: number analyzed (Participants) | 387 | 400 | 49
  Fasting Glucose (mmol/L) - Low, Gr. 2 | 9 | 9 | 0
  Fasting Glucose (mmol/L) - Low, Gr. 3: number analyzed (Participants) | 387 | 400 | 49
  Fasting Glucose (mmol/L) - Low, Gr. 3 | 1 | 2 | 0
  Fasting Glucose (mmol/L) - Low, Gr. 4: number analyzed (Participants) | 387 | 400 | 49
  Fasting Glucose (mmol/L) - Low, Gr. 4 | 0 | 3 | 2
  Fasting Glucose (mmol/L) - High, Any Gr.: number analyzed (Participants) | 387 | 400 | 49
  Fasting Glucose (mmol/L) - High, Any Gr. | 271 | 299 | 34
  Fasting Glucose (mmol/L) - High, Gr. 1: number analyzed (Participants) | 387 | 400 | 49
  Fasting Glucose (mmol/L) - High, Gr. 1 | 168 | 192 | 26
  Fasting Glucose (mmol/L) - High, Gr. 2: number analyzed (Participants) | 387 | 400 | 49
  Fasting Glucose (mmol/L) - High, Gr. 2 | 83 | 78 | 8
  Fasting Glucose (mmol/L) - High, Gr. 3: number analyzed (Participants) | 387 | 400 | 49
  Fasting Glucose (mmol/L) - High, Gr. 3 | 20 | 26 | 0
  Fasting Glucose (mmol/L) - High, Gr. 4: number analyzed (Participants) | 387 | 400 | 49
  Fasting Glucose (mmol/L) - High, Gr. 4 | 0 | 3 | 0
  GGT (U/L) - High, Any Gr.: number analyzed (Participants) | 375 | 394 | 48
  GGT (U/L) - High, Any Gr. | 209 | 225 | 14
  GGT (U/L) - High, Gr. 1: number analyzed (Participants) | 375 | 394 | 48
  GGT (U/L) - High, Gr. 1 | 133 | 144 | 9
  GGT (U/L) - High, Gr. 2: number analyzed (Participants) | 375 | 394 | 48
  GGT (U/L) - High, Gr. 2 | 41 | 52 | 4
  GGT (U/L) - High, Gr. 3: number analyzed (Participants) | 375 | 394 | 48
  GGT (U/L) - High, Gr. 3 | 30 | 27 | 1
  GGT (U/L) - High, Gr. 4: number analyzed (Participants) | 375 | 394 | 48
  GGT (U/L) - High, Gr. 4 | 5 | 2 | 0
  Magnesium (mmol/L) - Low, Any Gr.: number analyzed (Participants) | 371 | 398 | 49
  Magnesium (mmol/L) - Low, Any Gr. | 79 | 117 | 8
  Magnesium (mmol/L) - Low, Gr. 1: number analyzed (Participants) | 371 | 398 | 49
  Magnesium (mmol/L) - Low, Gr. 1 | 71 | 98 | 6
  Magnesium (mmol/L) - Low, Gr. 2: number analyzed (Participants) | 371 | 398 | 49
  Magnesium (mmol/L) - Low, Gr. 2 | 7 | 13 | 0
  Magnesium (mmol/L) - Low, Gr. 3: number analyzed (Participants) | 371 | 398 | 49
  Magnesium (mmol/L) - Low, Gr. 3 | 1 | 3 | 0
  Magnesium (mmol/L) - Low, Gr. 4: number analyzed (Participants) | 371 | 398 | 49
  Magnesium (mmol/L) - Low, Gr. 4 | 0 | 3 | 2
  Magnesium (mmol/L) - High, Any Gr.: number analyzed (Participants) | 371 | 398 | 49
  Magnesium (mmol/L) - High, Any Gr. | 76 | 105 | 16
  Magnesium (mmol/L) - High, Gr. 1: number analyzed (Participants) | 371 | 398 | 49
  Magnesium (mmol/L) - High, Gr. 1 | 58 | 80 | 11
  Magnesium (mmol/L) - High, Gr. 2: number analyzed (Participants) | 371 | 398 | 49
  Magnesium (mmol/L) - High, Gr. 2 | 0 | 0 | 0
  Magnesium (mmol/L) - High, Gr. 3: number analyzed (Participants) | 371 | 398 | 49
  Magnesium (mmol/L) - High, Gr. 3 | 18 | 22 | 4
  Magnesium (mmol/L) - High, Gr. 4: number analyzed (Participants) | 371 | 398 | 49
  Magnesium (mmol/L) - High, Gr. 4 | 0 | 3 | 1
  Potassium (mmol/L) - Low, Any Gr.: number analyzed (Participants) | 389 | 401 | 49
  Potassium (mmol/L) - Low, Any Gr. | 80 | 144 | 11
  Potassium (mmol/L) - Low, Gr. 1: number analyzed (Participants) | 389 | 401 | 49
  Potassium (mmol/L) - Low, Gr. 1 | 0 | 0 | 0
  Potassium (mmol/L) - Low, Gr. 2: number analyzed (Participants) | 389 | 401 | 49
  Potassium (mmol/L) - Low, Gr. 2 | 68 | 118 | 8
  Potassium (mmol/L) - Low, Gr. 3: number analyzed (Participants) | 389 | 401 | 49
  Potassium (mmol/L) - Low, Gr. 3 | 10 | 18 | 2
  Potassium (mmol/L) - Low, Gr. 4: number analyzed (Participants) | 389 | 401 | 49
  Potassium (mmol/L) - Low, Gr. 4 | 2 | 8 | 1
  Potassium (mmol/L) - High, Any Gr.: number analyzed (Participants) | 389 | 401 | 49
  Potassium (mmol/L) - High, Any Gr. | 67 | 78 | 13
  Potassium (mmol/L) - High, Gr. 1: number analyzed (Participants) | 389 | 401 | 49
  Potassium (mmol/L) - High, Gr. 1 | 49 | 55 | 11
  Potassium (mmol/L) - High, Gr. 2: number analyzed (Participants) | 389 | 401 | 49
  Potassium (mmol/L) - High, Gr. 2 | 15 | 17 | 2
  Potassium (mmol/L) - High, Gr. 3: number analyzed (Participants) | 389 | 401 | 49
  Potassium (mmol/L) - High, Gr. 3 | 3 | 6 | 0
  Potassium (mmol/L) - High, Gr. 4: number analyzed (Participants) | 389 | 401 | 49
  Potassium (mmol/L) - High, Gr. 4 | 0 | 0 | 0
  SGOT (U/L) - High, Any Gr.: number analyzed (Participants) | 389 | 400 | 49
  SGOT (U/L) - High, Any Gr. | 184 | 193 | 17
  SGOT (U/L) - High, Gr. 1: number analyzed (Participants) | 389 | 400 | 49
  SGOT (U/L) - High, Gr. 1 | 169 | 170 | 15
  SGOT (U/L) - High, Gr. 2: number analyzed (Participants) | 389 | 400 | 49
  SGOT (U/L) - High, Gr. 2 | 11 | 12 | 2
  SGOT (U/L) - High, Gr. 3: number analyzed (Participants) | 389 | 400 | 49
  SGOT (U/L) - High, Gr. 3 | 4 | 10 | 0
  SGOT (U/L) - High, Gr. 4: number analyzed (Participants) | 389 | 400 | 49
  SGOT (U/L) - High, Gr. 4 | 0 | 1 | 0
  SGPT (U/L) - High, Any Gr.: number analyzed (Participants) | 390 | 400 | 49
  SGPT (U/L) - High, Any Gr. | 195 | 209 | 19
  SGPT (U/L) - High, Gr. 1: number analyzed (Participants) | 390 | 400 | 49
  SGPT (U/L) - High, Gr. 1 | 172 | 175 | 17
  SGPT (U/L) - High, Gr. 2: number analyzed (Participants) | 390 | 400 | 49
  SGPT (U/L) - High, Gr. 2 | 18 | 19 | 2
  SGPT (U/L) - High, Gr. 3: number analyzed (Participants) | 390 | 400 | 49
  SGPT (U/L) - High, Gr. 3 | 5 | 14 | 0
  SGPT (U/L) - High, Gr. 4: number analyzed (Participants) | 390 | 400 | 49
  SGPT (U/L) - High, Gr. 4 | 0 | 1 | 0
  Sodium (mmol/L) - Low, Any Gr.: number analyzed (Participants) | 389 | 402 | 49
  Sodium (mmol/L) - Low, Any Gr. | 109 | 135 | 25
  Sodium (mmol/L) - Low, Gr. 1: number analyzed (Participants) | 389 | 402 | 49
  Sodium (mmol/L) - Low, Gr. 1 | 87 | 121 | 22
  Sodium (mmol/L) - Low, Gr. 2: number analyzed (Participants) | 389 | 402 | 49
  Sodium (mmol/L) - Low, Gr. 2 | 0 | 0 | 0
  Sodium (mmol/L) - Low, Gr. 3: number analyzed (Participants) | 389 | 402 | 49
  Sodium (mmol/L) - Low, Gr. 3 | 21 | 12 | 1
  Sodium (mmol/L) - Low, Gr. 4: number analyzed (Participants) | 389 | 402 | 49
  Sodium (mmol/L) - Low, Gr. 4 | 1 | 2 | 2
  Sodium (mmol/L) - High, Any Gr.: number analyzed (Participants) | 389 | 402 | 49
  Sodium (mmol/L) - High, Any Gr. | 76 | 103 | 9
  Sodium (mmol/L) - High, Gr. 1: number analyzed (Participants) | 389 | 402 | 49
  Sodium (mmol/L) - High, Gr. 1 | 71 | 91 | 7
  Sodium (mmol/L) - High, Gr. 2: number analyzed (Participants) | 389 | 402 | 49
  Sodium (mmol/L) - High, Gr. 2 | 4 | 9 | 2
  Sodium (mmol/L) - High, Gr. 3: number analyzed (Participants) | 389 | 402 | 49
  Sodium (mmol/L) - High, Gr. 3 | 1 | 2 | 0
  Sodium (mmol/L) - High, Gr. 4: number analyzed (Participants) | 389 | 402 | 49
  Sodium (mmol/L) - High, Gr. 4 | 0 | 1 | 0
  Total Bilirubin (umol/L) - High, Any Gr.: number analyzed (Participants) | 390 | 401 | 49
  Total Bilirubin (umol/L) - High, Any Gr. | 35 | 57 | 7
  Total Bilirubin (umol/L) - High, Gr. 1: number analyzed (Participants) | 390 | 401 | 49
  Total Bilirubin (umol/L) - High, Gr. 1 | 26 | 44 | 6
  Total Bilirubin (umol/L) - High, Gr. 2: number analyzed (Participants) | 390 | 401 | 49
  Total Bilirubin (umol/L) - High, Gr. 2 | 7 | 9 | 0
  Total Bilirubin (umol/L) - High, Gr. 3: number analyzed (Participants) | 390 | 401 | 49
  Total Bilirubin (umol/L) - High, Gr. 3 | 2 | 2 | 0
  Total Bilirubin (umol/L) - High, Gr. 4: number analyzed (Participants) | 390 | 401 | 49
  Total Bilirubin (umol/L) - High, Gr. 4 | 0 | 2 | 1
  Uric Acid (umol/L) - High, Any Gr.: number analyzed (Participants) | 370 | 397 | 49
  Uric Acid (umol/L) - High, Any Gr. | 118 | 113 | 15
  Uric Acid (umol/L) - High, Gr. 1: number analyzed (Participants) | 370 | 397 | 49
  Uric Acid (umol/L) - High, Gr. 1 | 0 | 0 | 0
  Uric Acid (umol/L) - High, Gr. 2: number analyzed (Participants) | 370 | 397 | 49
  Uric Acid (umol/L) - High, Gr. 2 | 0 | 0 | 0
  Uric Acid (umol/L) - High, Gr. 3: number analyzed (Participants) | 370 | 397 | 49
  Uric Acid (umol/L) - High, Gr. 3 | 116 | 98 | 10
  Uric Acid (umol/L) - High, Gr. 4: number analyzed (Participants) | 370 | 397 | 49
  Uric Acid (umol/L) - High, Gr. 4 | 2 | 15 | 5

17. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Hematology Tests by Highest Grade According to NCI-CTCAE v3.0 During the Treatment Period
Description: Clinical laboratory tests for hematology parameters were performed at local laboratories; any abnormal values (High or Low) were based on local laboratory normal ranges. Laboratory abnormalities are presented by the highest grade according to NCI-CTCAE v3.0. Not every abnormal laboratory value qualified as an adverse event, only if it met any of the following criteria: clinically significant (per investigator); accompanied by clinical symptoms; resulted in a change in study treatment; or required a change in concomitant therapy. Median [range] time on study treatment per arm: Placebo: 49.3 [0.3-514.7] weeks; Pertuzumab: 75.7 [0.6-519.6] weeks; Crossover: 129.9 [0.3-322.3] weeks. INR = International Normalized Ratio; PTT = partial thromboplastin time; WBC = white blood cell
Time Frame: On Day 1 (and Day 8 for some measures) of every treatment cycle (1 cycle is 21 days) until Treatment Discontinuation Visit (see Description for time on study treatment per arm)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Trastuzumab + Docetaxel | Pertuzumab + Trastuzumab + Docetaxel | Crossover From Placebo to Pertuzumab
Number analyzed (Participants) | 396 | 408 | 50
Participants
  Hemoglobin (g/L) - Low, Any Grade (Gr.): number analyzed (Participants) | 392 | 404 | 49
  Hemoglobin (g/L) - Low, Any Grade (Gr.) | 350 | 372 | 20
  Hemoglobin (g/L) - Low, Gr. 1: number analyzed (Participants) | 392 | 404 | 49
  Hemoglobin (g/L) - Low, Gr. 1 | 202 | 186 | 9
  Hemoglobin (g/L) - Low, Gr. 2: number analyzed (Participants) | 392 | 404 | 49
  Hemoglobin (g/L) - Low, Gr. 2 | 127 | 161 | 6
  Hemoglobin (g/L) - Low, Gr. 3: number analyzed (Participants) | 392 | 404 | 49
  Hemoglobin (g/L) - Low, Gr. 3 | 21 | 25 | 5
  Hemoglobin (g/L) - Low, Gr. 4: number analyzed (Participants) | 392 | 404 | 49
  Hemoglobin (g/L) - Low, Gr. 4 | 0 | 0 | 0
  Hemoglobin (g/L) - High, Any Gr.: number analyzed (Participants) | 392 | 404 | 49
  Hemoglobin (g/L) - High, Any Gr. | 10 | 23 | 4
  Hemoglobin (g/L) - High, Gr. 1: number analyzed (Participants) | 392 | 404 | 49
  Hemoglobin (g/L) - High, Gr. 1 | 9 | 20 | 2
  Hemoglobin (g/L) - High, Gr. 2: number analyzed (Participants) | 392 | 404 | 49
  Hemoglobin (g/L) - High, Gr. 2 | 1 | 2 | 0
  Hemoglobin (g/L) - High, Gr. 3: number analyzed (Participants) | 392 | 404 | 49
  Hemoglobin (g/L) - High, Gr. 3 | 0 | 1 | 2
  Hemoglobin (g/L) - High, Gr. 4: number analyzed (Participants) | 392 | 404 | 49
  Hemoglobin (g/L) - High, Gr. 4 | 0 | 0 | 0
  Lymphocytes (10^9/L) - Low, Any Gr.: number analyzed (Participants) | 391 | 404 | 49
  Lymphocytes (10^9/L) - Low, Any Gr. | 259 | 276 | 8
  Lymphocytes (10^9/L) - Low, Gr. 1: number analyzed (Participants) | 391 | 404 | 49
  Lymphocytes (10^9/L) - Low, Gr. 1 | 36 | 39 | 0
  Lymphocytes (10^9/L) - Low, Gr. 2: number analyzed (Participants) | 391 | 404 | 49
  Lymphocytes (10^9/L) - Low, Gr. 2 | 128 | 136 | 4
  Lymphocytes (10^9/L) - Low, Gr. 3: number analyzed (Participants) | 391 | 404 | 49
  Lymphocytes (10^9/L) - Low, Gr. 3 | 64 | 69 | 3
  Lymphocytes (10^9/L) - Low, Gr. 4: number analyzed (Participants) | 391 | 404 | 49
  Lymphocytes (10^9/L) - Low, Gr. 4 | 31 | 32 | 1
  Lymphocytes (10^9/L)- High, Any Gr.: number analyzed (Participants) | 391 | 404 | 49
  Lymphocytes (10^9/L)- High, Any Gr. | 58 | 72 | 9
  Lymphocytes (10^9/L)- High, Gr. 1: number analyzed (Participants) | 391 | 404 | 49
  Lymphocytes (10^9/L)- High, Gr. 1 | 0 | 0 | 0
  Lymphocytes (10^9/L)- High, Gr. 2: number analyzed (Participants) | 391 | 404 | 49
  Lymphocytes (10^9/L)- High, Gr. 2 | 49 | 57 | 6
  Lymphocytes (10^9/L)- High, Gr. 3: number analyzed (Participants) | 391 | 404 | 49
  Lymphocytes (10^9/L)- High, Gr. 3 | 9 | 15 | 3
  Lymphocytes (10^9/L)- High, Gr. 4: number analyzed (Participants) | 391 | 404 | 49
  Lymphocytes (10^9/L)- High, Gr. 4 | 0 | 0 | 0
  Neutrophils (10^9/L)- Low, Any Gr.: number analyzed (Participants) | 391 | 404 | 49
  Neutrophils (10^9/L)- Low, Any Gr. | 349 | 371 | 2
  Neutrophils (10^9/L)- Low, Gr. 1: number analyzed (Participants) | 391 | 404 | 49
  Neutrophils (10^9/L)- Low, Gr. 1 | 7 | 4 | 0
  Neutrophils (10^9/L)- Low, Gr. 2: number analyzed (Participants) | 391 | 404 | 49
  Neutrophils (10^9/L)- Low, Gr. 2 | 25 | 34 | 0
  Neutrophils (10^9/L)- Low, Gr. 3: number analyzed (Participants) | 391 | 404 | 49
  Neutrophils (10^9/L)- Low, Gr. 3 | 81 | 99 | 0
  Neutrophils (10^9/L)- Low, Gr. 4: number analyzed (Participants) | 391 | 404 | 49
  Neutrophils (10^9/L)- Low, Gr. 4 | 236 | 234 | 2
  PTT (sec) - High, Any Gr.: number analyzed (Participants) | 28 | 35 | 3
  PTT (sec) - High, Any Gr. | 6 | 9 | 1
  PTT (sec) - High, Gr. 1: number analyzed (Participants) | 28 | 35 | 3
  PTT (sec) - High, Gr. 1 | 5 | 2 | 1
  PTT (sec) - High, Gr. 2: number analyzed (Participants) | 28 | 35 | 3
  PTT (sec) - High, Gr. 2 | 0 | 4 | 0
  PTT (sec) - High, Gr. 3: number analyzed (Participants) | 28 | 35 | 3
  PTT (sec) - High, Gr. 3 | 1 | 3 | 0
  PTT (sec) - High, Gr. 4: number analyzed (Participants) | 28 | 35 | 3
  PTT (sec) - High, Gr. 4 | 0 | 0 | 0
  Platelets (10^9/L) - Low, Any Gr.: number analyzed (Participants) | 392 | 404 | 49
  Platelets (10^9/L) - Low, Any Gr. | 82 | 92 | 13
  Platelets (10^9/L) - Low, Gr. 1: number analyzed (Participants) | 392 | 404 | 49
  Platelets (10^9/L) - Low, Gr. 1 | 75 | 78 | 11
  Platelets (10^9/L) - Low, Gr. 2: number analyzed (Participants) | 392 | 404 | 49
  Platelets (10^9/L) - Low, Gr. 2 | 5 | 5 | 0
  Platelets (10^9/L) - Low, Gr. 3: number analyzed (Participants) | 392 | 404 | 49
  Platelets (10^9/L) - Low, Gr. 3 | 2 | 3 | 0
  Platelets (10^9/L) - Low, Gr. 4: number analyzed (Participants) | 392 | 404 | 49
  Platelets (10^9/L) - Low, Gr. 4 | 0 | 6 | 2
  Prothrombin Time (INR) - High, Any Gr.: number analyzed (Participants) | 198 | 216 | 14
  Prothrombin Time (INR) - High, Any Gr. | 135 | 157 | 11
  Prothrombin Time (INR) - High, Gr. 1: number analyzed (Participants) | 198 | 216 | 14
  Prothrombin Time (INR) - High, Gr. 1 | 127 | 136 | 9
  Prothrombin Time (INR) - High, Gr. 2: number analyzed (Participants) | 198 | 216 | 14
  Prothrombin Time (INR) - High, Gr. 2 | 3 | 6 | 0
  Prothrombin Time (INR) - High, Gr. 3: number analyzed (Participants) | 198 | 216 | 14
  Prothrombin Time (INR) - High, Gr. 3 | 5 | 15 | 2
  Prothrombin Time (INR) - High, Gr. 4: number analyzed (Participants) | 198 | 216 | 14
  Prothrombin Time (INR) - High, Gr. 4 | 0 | 0 | 0
  WBC (10^9/L) - Low, Any Gr.: number analyzed (Participants) | 392 | 404 | 49
  WBC (10^9/L) - Low, Any Gr. | 366 | 387 | 5
  WBC (10^9/L) - Low, Gr. 1: number analyzed (Participants) | 392 | 404 | 49
  WBC (10^9/L) - Low, Gr. 1 | 36 | 34 | 1
  WBC (10^9/L) - Low, Gr. 2: number analyzed (Participants) | 392 | 404 | 49
  WBC (10^9/L) - Low, Gr. 2 | 92 | 92 | 3
  WBC (10^9/L) - Low, Gr. 3: number analyzed (Participants) | 392 | 404 | 49
  WBC (10^9/L) - Low, Gr. 3 | 186 | 206 | 0
  WBC (10^9/L) - Low, Gr. 4: number analyzed (Participants) | 392 | 404 | 49
  WBC (10^9/L) - Low, Gr. 4 | 52 | 55 | 1
  WBC (10^9/L) - High, Any Gr.: number analyzed (Participants) | 392 | 404 | 49
  WBC (10^9/L) - High, Any Gr. | 0 | 3 | 1
  WBC (10^9/L) - High, Gr. 1: number analyzed (Participants) | 392 | 404 | 49
  WBC (10^9/L) - High, Gr. 1 | 0 | 0 | 0
  WBC (10^9/L) - High, Gr. 2: number analyzed (Participants) | 392 | 404 | 49
  WBC (10^9/L) - High, Gr. 2 | 0 | 0 | 0
  WBC (10^9/L) - High, Gr. 3: number analyzed (Participants) | 392 | 404 | 49
  WBC (10^9/L) - High, Gr. 3 | 0 | 3 | 1
  WBC (10^9/L) - High, Gr. 4: number analyzed (Participants) | 392 | 404 | 49
  WBC (10^9/L) - High, Gr. 4 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first treatment dose (12-Feb-2008) through to end of study (23-Nov-2018) for a total safety analysis timeframe of 10 years, 9.5 months.
Description: Of enrolled participants (Pertuzumab [Ptz]: N=402, Placebo [Pla]: N=406), 2 in each arm received no treatment (total of 4), 9 in Pla arm received at least 1 dose of Ptz, and 1 in Ptz arm received Pla at every cycle; resulting in a Safety Population of Ptz: N=408 (402-2+9-1), Pla: N=396 (406-2-9+1), and 50 participants in Pla arm crossed over to Ptz.
Arm/Group | Placebo + Trastuzumab + Docetaxel | Pertuzumab + Trastuzumab + Docetaxel | Crossover From Placebo to Pertuzumab
All-Cause Mortality (participants affected / at risk) | 261/396 | 238/408 | 14/50
Serious Adverse Events (participants affected / at risk) | 116/396 | 160/408 | 10/50
Other Adverse Events (participants affected / at risk) | 386/396 | 400/408 | 45/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Trastuzumab + Docetaxel (N=396) | Pertuzumab + Trastuzumab + Docetaxel (N=408) | Crossover From Placebo to Pertuzumab (N=50)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (4) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 20 (23) | 46 (48) | 0 (0)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 19 (20) | 18 (23) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 7 (7) | 6 (6) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 13 (16) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Drowning (General disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 6 (6) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 3 (3) | 3 (3) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 3 (3) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 10 (12) | 0 (0)
Cellulitis gangrenous (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Coccidioidomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (3) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
H1N1 influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Lymph node tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neutropenic infection (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 11 (11) | 7 (7) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood electrolytes abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Breast haemorrhage (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (5) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Trastuzumab + Docetaxel (N=396) | Pertuzumab + Trastuzumab + Docetaxel (N=408) | Crossover From Placebo to Pertuzumab (N=50)
Fatigue (General disorders) | 148 (291) | 156 (320) | 5 (16)
Asthenia (General disorders) | 122 (268) | 114 (265) | 3 (3)
Oedema peripheral (General disorders) | 111 (163) | 102 (141) | 1 (1)
Mucosal inflammation (General disorders) | 78 (111) | 111 (185) | 1 (1)
Pyrexia (General disorders) | 72 (94) | 81 (138) | 3 (6)
Oedema (General disorders) | 49 (76) | 49 (84) | 1 (1)
Chills (General disorders) | 15 (18) | 34 (36) | 1 (7)
Pain (General disorders) | 22 (26) | 26 (31) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 191 (428) | 277 (989) | 25 (155)
Nausea (Gastrointestinal disorders) | 168 (359) | 184 (394) | 4 (7)
Vomiting (Gastrointestinal disorders) | 96 (150) | 110 (184) | 5 (7)
Constipation (Gastrointestinal disorders) | 100 (179) | 69 (135) | 4 (6)
Stomatitis (Gastrointestinal disorders) | 63 (138) | 82 (167) | 6 (13)
Abdominal pain (Gastrointestinal disorders) | 50 (66) | 64 (86) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 48 (73) | 55 (80) | 3 (8)
Abdominal pain upper (Gastrointestinal disorders) | 43 (54) | 44 (69) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 240 (256) | 248 (264) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 96 (185) | 156 (288) | 11 (19)
Nail disorder (Skin and subcutaneous tissue disorders) | 92 (105) | 96 (106) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 40 (67) | 75 (117) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 25 (26) | 47 (53) | 4 (6)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 22 (25) | 28 (38) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 20 (27) | 23 (28) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 191 (797) | 209 (849) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 77 (143) | 100 (151) | 6 (15)
Leukopenia (Blood and lymphatic system disorders) | 82 (344) | 75 (288) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 79 (114) | 95 (138) | 1 (1)
Headache (Nervous system disorders) | 76 (128) | 106 (187) | 7 (9)
Dysgeusia (Nervous system disorders) | 62 (116) | 75 (95) | 1 (30)
Peripheral sensory neuropathy (Nervous system disorders) | 59 (82) | 52 (93) | 2 (2)
Dizziness (Nervous system disorders) | 53 (73) | 67 (133) | 4 (4)
Paraesthesia (Nervous system disorders) | 41 (60) | 43 (52) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 98 (209) | 97 (202) | 5 (30)
Arthralgia (Musculoskeletal and connective tissue disorders) | 71 (130) | 83 (133) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 52 (79) | 76 (116) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 48 (58) | 66 (98) | 6 (17)
Bone pain (Musculoskeletal and connective tissue disorders) | 31 (56) | 37 (48) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 38 (57) | 40 (51) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 20 (24) | 50 (94) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 79 (118) | 101 (146) | 6 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 62 (87) | 67 (99) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 35 (47) | 41 (56) | 2 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 27 (32) | 32 (55) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 23 (29) | 33 (43) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 106 (176) | 120 (229) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 21 (28) | 37 (60) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 57 (99) | 90 (174) | 13 (32)
Nasopharyngitis (Infections and infestations) | 60 (108) | 76 (161) | 13 (58)
Urinary tract infection (Infections and infestations) | 29 (39) | 39 (65) | 4 (6)
Paronychia (Infections and infestations) | 16 (23) | 32 (45) | 6 (8)
Lacrimation increased (Eye disorders) | 55 (63) | 60 (74) | 0 (0)
Conjunctivitis (Infections and infestations) | 19 (22) | 31 (45) | 2 (2)
Insomnia (Psychiatric disorders) | 55 (72) | 67 (95) | 2 (3)
Depression (Psychiatric disorders) | 20 (22) | 26 (33) | 2 (2)
Hypertension (Vascular disorders) | 31 (93) | 53 (83) | 4 (4)
Hot flush (Vascular disorders) | 21 (39) | 23 (26) | 0 (0)
Weight decreased (Investigations) | 19 (22) | 37 (51) | 3 (3)
Weight increased (Investigations) | 22 (35) | 17 (21) | 0 (0)
Hypersensitivity (Immune system disorders) | 21 (29) | 28 (33) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 27 (33) | 27 (43) | 3 (9)
Dysuria (Renal and urinary disorders) | 11 (12) | 23 (27) | 0 (0)
Influenza (Infections and infestations) | 22 (33) | 30 (43) | 6 (10)
Rhinitis (Infections and infestations) | 22 (35) | 22 (50) | 4 (13)
Dry eye (Eye disorders) | 8 (8) | 24 (27) | 2 (2)
Anxiety (Psychiatric disorders) | 20 (28) | 20 (25) | 1 (1)
Lymphoedema (Vascular disorders) | 16 (18) | 24 (25) | 0 (0)
Chest pain (General disorders) | 21 (24) | 15 (17) | 0 (0)
Influenza like illness (General disorders) | 10 (12) | 23 (41) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 7 (8) | 3 (3)
Gastritis (Gastrointestinal disorders) | 7 (8) | 16 (20) | 3 (3)
Pneumonia (Infections and infestations) | 8 (8) | 12 (20) | 4 (4)
Cystitis (Infections and infestations) | 6 (7) | 16 (25) | 5 (6)
Cellulitis (Infections and infestations) | 12 (14) | 16 (20) | 3 (6)
Bronchitis (Infections and infestations) | 15 (19) | 16 (29) | 4 (5)
Pharyngitis (Infections and infestations) | 9 (10) | 22 (28) | 3 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (24) | 17 (19) | 3 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 17 (22) | 22 (27) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 5 (6) | 5 (5) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 11 (15) | 21 (28) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.